

# Statistical Analysis Plan

NCT Number: NCT03706456

Title: A Phase 3, Multicenter, Open-Label, Uncontrolled Study to Evaluate the Efficacy and Safety of Cx601 in the Treatment of Complex Perianal Fistulas in Adult Patients with Crohn's Disease

Study Number: Darvadstrocel-3002

Document Version and Date

Analysis using Data up to Week 24: Version 2 / 02-Sep-2020 Analysis using Data up to Week 52: Version 2 / 05-Mar-2021 Analysis using Data up to Week 156: Version 1 / 09-May-2022

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.



# STATISTICAL ANALYSIS PLAN

[Analysis using Data up to Week 24]

STUDY NUMBER: Darvadstrocel-3002

the applicable terms of Use the Eff A Phase 3, Multicenter, Open-Label, Uncontrolled Study to Evaluate the Efficacy and Safety of Cx601 in the Treatment of Complex Perianal Fistulas in Adult Patients with Crohn's Disease

Version: 2nd
Date: 2 September 2020

Prepared by:

Based on:

Protocol Version: Amendment 3

Property of Lakeda. Protocol Date: 9 October 2019

Property of Takeda. For non-commercial use only and subject to the applicable Tames of use

# 2.0 TABLE OF CONTENTS

| 1.0 | TITLE | E PAGE | |
|---|---|---|---|
| 1. | 1 <b>A</b> p | pproval Signatures | |
| 2.0 | TABL | E OF CONTENTS | |
| Li | st of In- | Text Tables | |
| Li | st of In- | Text Figures | <u>≥</u> <sup>∠</sup> |
| 3.0 | LIST | OF ABBREVIATIONS | 4 |
| 4.0 | OBJE | OF ABBREVIATIONS. CTIVES. imary Objectives. | <i>(</i> |
| 4. | 1 Pr | imary Objectives | <i>6</i> |
| 4. | 2 Se | condary Objectives | <i>6</i> |
| 4 | 3 Ad | lditional Objectives | <i>6</i> |
| 4.4 | 4 St | ıdy Design | <i>6</i> |
| 5.0 | ANAI | LYSIS ENDPOINTS | 8 |
| 5. | 1 Pr | imary Endpoint | 8 |
| 5 | 2 Se | condary Endpoints | 8 |
| 5 | 3 Sa | fety Endpoints | 9 |
| 5.4 | 4 Ac | lditional Endpoints | 9 |
| 6.0 | DETE | condary Objectives Iditional Objectives Idy Design LYSIS ENDPOINTS Imary Endpoint condary Endpoints fety Endpoints Iditional Endpoints RMINATION OF SAMPLE SIZE | 10 |
| 7.0 | IVIE I F | ODS OF ANALYSIS AND PRESENTATION | 1 1 |
| 7. | 1 Ge | Study Definitions Study Definitions | 11 |
| | 7.1.1 | | |
| | 7.1.2 | Definition of Study Days | |
| | 7.1.3 | Definition of Study Visit Windows | |
| | 7.1.4 | Significance Devel and Confidence Coefficient. | 16 |
| | 7.1.5 | Calculation of Combined Remission, Clinical Remission, Response | |
| | 7.1.6 | Calculation of Relapse in Subjects with Clinical/Combined Remission | 17 |
| 7.3 | | alysis Sets | |
| 7. | 3 Di | sposition of Subjects | |
| | 737 | Study Information | |
| 1 | 7.3.2 | Screen Failures | |
| (1) | 7.3.3 | Subject Eligibility | |
| | 7.3.4 | Number of Subjects Who Entered the Treatment Period by Site | |
| | 7.3.5 | Disposition of Subjects for Follow-up Period. | |
| | 7.3.6 | Completion Status for Follow-up Period | |
| | 737 | Disposition of Subjects for Long-Term Follow-up Period | 21 |

Figure 4.a

| 7.3.8 | Completion Status for Long-Term Follow-up Period | 22 |
|---|---|---|
| 7.3.9 | | |
| 7.4 D | emographic and Other Baseline Characteristics | 24 |
| | fedical History and Concurrent Medical Conditions | |
| 7.6 M | fedication History and Concomitant Medications | 25 |
| 7.7 St | tudy Drug Exposure and Compliance | 2 <i>6</i> |
| 7.8 E | fficacy Analysis | 2 <i>e</i> |
| 7.8.1 | tudy Drug Exposure and Compliance fficacy Analysis Primary Endpoint Secondary Endpoints Additional Endpoints Statistical/Analytical Issues | 27 |
| 7.8.2 | Secondary Endpoints | 27 |
| 7.8.3 | Additional Endpoints | 30 |
| 7.8.4 | Statistical/Analytical Issues | 31 |
| 7.9 O | ther Outcomes | 32 |
| 7.10 Sa | afety Analysis | 32 |
| 7.10.1 | Statistical/Analytical Issues ther Outcomes afety Analysis | 33 |
| 7.10.2 | 2 Clinical Laboratory Evaluations | 37 |
| 7.10.3 | 3 Vital Signs | 39 |
| 7.10.4 | 4 Other Observations Related to Safety | 39 |
| 7.11 In | nterim Analysis | 41 |
| 8.0 REFE | ERENCES | 52 |
| 9.0 APPE | ENDIX | 53 |
| LIST OF IN | -TEXT TABLES | |
| Table 7.a | Visit Window of Fistula MRI Assessment | 13 |
| Table 7.b | Visit Window of Fistula Clinical Assessment | |
| Table 7.c | Visit Window of PDAI Score | |
| Table 7.d | Visit Window of CDAI Score | |
| Table 7.e | Visit Window of Van Assche Score | |
| Table 7.6 | Visit Window of Vital Signs | |
| Table 7.g | Visit Window of Clinical Laboratory Tests | |
| Table 7.h | Visit Window of Anti-donor Antibody Test | |
| J. | | |
| I ICT OF IN | TEVT FICTIDES | |

#### 3.0 LIST OF ABBREVIATIONS

AΕ adverse event

ALP alkaline phosphatase ALT alanine aminotransferase AST aspartate aminotransferase **CDAI** Crohn's Disease Activity Index **DMEM** Dulbecco Modified Eagle's Medium

eASC expanded allogeneic adipose-derived stem cells

**ECG** electrocardiogram

eCRF electronic case report form **EMA** European Medicines Agency

EO **External Opening** 

**FDA** Food and Drug Administration

**GCP** Good Clinical Practice

**GGT** gamma-glutamyl transpeptidase hepatitis B virus surface antigen HBsAg

**HBV** hepatitis B virus

hCG human chorionic gonadotropin

**HCV** hepatitis C virus **HSA** human serum albumin

International Conference on Harmonisation **ICH** 

ILinterleukin

international normalized ratio INR

Ю Internal Opening institutional review board IRB

intention to treat ITT

LOCF last observation carried forward

Medical Dictionary for Regulatory Activities MedDRA **MHLW** Ministry of Health, Labour and Welfare

Medicines and Healthcare products Regulatory Agency **MHRA** 

'akedai. For non' modified intention to treat mITT MRI magnetic resonance imaging PCR polymerase chain reaction PDAI Perianal Disease Activity Index

**PMDA** Pharmaceuticals and Medical Devices Agency

PPS per protocol set PTE Pretreatment event SAE serious adverse event SAP statistical analysis plan

SUSAR suspected unexpected serious adverse reaction

TEAE treatment-emergent AE TNF tumor necrosis factor ULN upper limit of normal **WBC** white blood cell

# 4.0 OBJECTIVES

# 4.1 Primary Objectives

• To evaluate the efficacy of Cx601 for the treatment of complex perianal fistulas in adult patients with Crohn's disease over 24 weeks.

# 4.2 Secondary Objectives

- To evaluate the efficacy of Cx601 for the treatment of complex perianal fistulas in adult patients with Crohn's disease over 52 weeks.
- To evaluate the safety of Cx601 for the treatment of perianal fistulas in adult patients with Crohn's disease over minimum 156 weeks.

# 4.3 Additional Objectives

- To evaluate the absence of clinically relevant alloreactivity.
- To evaluate the effects of Cx601 on Crohn's disease activity and quality of life.

# 4.4 Study Design

This is Phase 3, a multicenter, open-label, uncontrolled study to evaluate the efficacy and safety of Cx601 in the treatment of complex perianal fistulas in adult patients with Crohn's disease.

Subjects with Crohn's disease whose complex perianal fistulas were previously treated and refractory (inadequate response, loss of response or intolerance) to at least one of the following treatments: antibiotics, immunosuppressants or biologics (anti-TNFs, anti-integrin or anti-IL-12/23) will be included in the study. Note that those subjects who are refractory to antibiotics only will be must be less than 25% of all subjects enrolled.

The study will permit continuation of baseline treatments for Crohn's disease in an add-on design (ie, biologics, immunosuppressants, etc.) . A total of 20 subjects are planned to be enrolled, and study product, cell suspension containing  $120\times10^6$  cells of eASCs, will be intralesionally injected to all participants. Since this is the first study of Cx601 in Japanese subjects, the enrollment of at least the first 3 subjects will be adjusted not to be administered the study product at the same day.

This study consists of the screening period (approximately 5 weeks prior to study product administration, including the screening visit and the preparation visit), the treatment period (the day of study product administration), the follow-up period (approximately 52 weeks after study product administration), and the long-term follow-up period (from Week 52 to Week 156 or later; for a minimum of 104 weeks). Cx601 will be administrated once on Day 1, and the efficacy and safety of Cx601 will be mainly evaluated in the subsequent 52-week follow-up period. The primary endpoint will be evaluated at Week 24. Additionally, in the long-term follow-up period after Week 52, a safety follow-up evaluation will be performed for all subjects every 26 weeks (6 months) until Week 156 or later.

In the screening period, a screening visit (Visit 1) to determine a subject's eligibility is scheduled during the period from Day -39 to the day before preparation. All the subjects eligible by the screening will receive fistula curettage and seton placement under anesthesia at the preparation visit (Visit 2: Day -21, done no later than Day -14). Seton(s) placed will be removed on the day of study product administration (Visit 3: Day 1), just before the administration of the study product. Appropriate training for the preparation and the administration will be implemented to standardize the procedures between study sites.

The subjects who meet all the eligibility criteria will visit the study site on Day 1, and receive fistula curettage under anesthesia and an intralesional injection of cell suspension containing 120×10<sup>6</sup> cells of eASCs (Cx601). Thereafter, in follow-up period, the subjects will visit the study site for the clinical assessments including fistula closure at Weeks 2, 4, 8, 16, 24, 40 and 52. Radiological assessments (MRI) of fistula closure will also be performed at Weeks 24 and 52.

Additionally, in the long-term follow-up period, the safety follow-up will be performed on all the subjects (where possible) every 26 weeks (6 months) from a visit in Week 52 through Week 156. This study will be switched to a post-marketing clinical study if Cx601 is approved before the study completion.

A schematic study design is shown in Figure 4.a.

Figure 4.a **Schematic Study Design** 



#### 5.0 ANALYSIS ENDPOINTS

#### 5.1 **Primary Endpoint**

Proportion of subjects with combined remission at Week 24.

#### 5.2 **Secondary Endpoints**

# Efficacy analysis using data up to Week 24:

- Proportion of subjects with clinical remission at Week 24.
- Proportion of subjects with response at Week 24.
- Time to clinical remission by Week 24.
- Time to response by Week 24.
- to the applicable terms of Use linics. Proportion of subjects with relapse at Week 24 in subjects with clinical remission at previous visit.
- Time to relapse by Week 24 in subjects with clinical remission at previous visit.
- PDAI score (including total score, discharge sub-score and pain sub-score) up to Week 24.
- CDAI score up to Week 24.
- Van Assche score up to Week 24.

# Efficacy analysis using data up to Week 52.

- Proportion of subjects with combined remission at Week 52.
- Proportion of subjects with clinical remission at Week 52.
- Proportion of subjects with response at Week 52.
- Time to combined remission by Week 52.
- Time to clinical remission by Week 52.
- Time to response by Week 52.
- Proportion of subjects with relapse at Week 52 in subjects with combined remission at Week 24.
- Time to relapse by Week 52 in subjects with combined remission at Week 24.
- PDAI score (including total score, discharge sub-score and pain sub-score) up to Week 52.
- CDAI score up to Week 52.
- Van Assche score up to Week 52.

esults in esults in the applicable of the applic

# 7.0 METHODS OF ANALYSIS AND PRESENTATION

# 7.1 General Principles

# 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE): An adverse event whose date of onset occurs on or after receiving study treatment.
- Pretreatment event (PTE): Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to study treatment administration.
- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles.
- Duration of study after baseline (days): Date of last visit/contact date of study treatment administration + 1.
   If subject is ongoing, date of last visit/contact will be imputed by date of data cut off.
- Duration of follow-up after baseline by Week 24 (weeks): (Date of the latest fistula clinical assessment or the latest visit by Day 198 date of study treatment administration + 1)/7.
- Duration of Crohn's Disease (years): Date of informed consent date of Crohn's disease diagnosis.
   (If month of diagnosis is missing, month will be replaced with January. If day of diagnosis is missing, day will be replaced with I<sup>SI</sup>.)
- Combined remission: Defined as the clinically confirmed closure of all treated external openings that were draining at the screening despite gentle finger compression, and absence of collections >2 cm in the treated fistulas which is confirmed by the central MRI assessment (a collection >2 cm is considered as present if at least two out of the 3 dimensions centrally assessed are >2 cm in any of fistula tract).
- Clinical remission: Defined as the clinically confirmed closure of all treated external openings that were draining at the screening despite gentle finger compression.
- Response: Defined as the clinically confirmed closure of at least 50% of all treated external openings that were draining at the screening despite gentle finger compression. Note: Clinically confirmed closure of at least 50% is defined as 1 closure for subjects with 1 baseline external opening, 1 or 2 closures for subjects with 2 baseline external openings, and 2 or 3 closures for subjects with 3 baseline external openings.
- Relapse: Defined as the clinically confirmed reopening of any of the treated external openings with active drainage, or the development of a collection >2 cm in the treated fistulas confirmed by central MRI assessment

(a collection >2 cm is considered as present if at least two out of the 3 dimensions centrally

- remission/response (days): The time from the study
  remission/response is observed.
  For combined remission, date is the latest of fistula MRI assessment and fistula clinical assessment.

  Time to relapse (days): The time from the first visit which the first visit by which relapse is observed.

  (Time to relapse by the first visit which the first visit by which relapse is observed.)
- defined as "the time from the combined remission at Week 24 to the first visit by which relapse is observed.)
- Presence/Absence of donor specific antibody: Results for each post-baseline visit will be presence when at least one of donor specific antibody tests (Class I and/or Class II) is presence, otherwise results will be absence. A result at baseline will represent presence/absence of anti-HLA Class I and Class II antibody.
- CDAI total score: CDAI total score and body weight will be cut-off by -10, i.e. score below -10 will be treated as -10.

# 7.1.2 Definition of Study Days

The following definitions and calculation formulas will be used.

Study Day: The day before study treatment administration will be defined as Study Day -1 and the day of the study treatment administration will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the study treatment administration, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.

# 7.1.3 Definition of Study Visit Windows

When calculating Study Day relative to a reference date (ie, study treatment administration [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

# 7.1.3.1 Fistula Assessment

All evaluable data (ie, non-missing data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the largest Study Day will be used.

Table 7.a Visit Window of Fistula MRI Assessment

| | Scheduled Study Day | | Time Interval (days) | |
|---|---|---|---|---|
| Visit | (da | ys) | Study Day | |
| Baseline | Study Day: | Day Before<br>Preparation | - Day Before Preparation | |
| Week 24 | Study Day: | 169 | 2 - 198 | ベ |
| Week 52 | Study Day: | 365 | 199 - 448 | 5 |
| Week 104 | Study Day: | 729 | 449 - 812 | |
| Week 156 | Study Day: | 1093 | 813 - | |
| Week 24(LOCF) | Study Day: | | 2 - 198 | |
| Week 52(LOCF) | Study Day: | | 2 - 448 | |
| Week 104(LOCF) | Study Day: | | 2 812 | |
| Week 156(LOCF) | Study Day: | | × O 2 - | |

Table 7.b

| Study Day. | | |
|---|---|---|
| dow of Fistula C | Clinical Ass | sessment |
| Scheduled S | tudy Day | Time Interval (days) |
| (day | s) | Study Day |
| Study Day: | Day Before<br>Preparation | - Day Before Preparation |
| Study Day: | <sub>0</sub> 15 | 2 - 22 |
| Study Day: | 29 | 23 - 43 |
| Study Day: | 57 | 44 - 85 |
| Study Day | 113 | 86 - 141 |
| Study Day: | 169 | 142 - 198 |
| Study Day: | 281 | 199 - 323 |
| Study Day: | 365 | 324 - 448 |
| Study Day: | 729 | 449 - 812 |
| Study Day: | 1093 | 813 - |
| Study Day: | | 2 - 22 |
| Study Day: | | 2 - 43 |
| Study Day: | | 2 - 85 |
| Study Day: | | 2 - 141 |
| Study Day: | | 2 - 198 |
| Study Day: | | 2 - 323 |
| Study Day: | | 2 - 448 |
| Study Day: | | 2 - 812 |
| Study Day: | | 2 - |
| | Study Day: | Scheduled Study Day (days) Study Day: Day Before Preparation Study Day: 15 Study Day: 29 Study Day: 57 Study Day: 169 Study Day: 169 Study Day: 365 Study Day: 729 Study Day: 1093 Study Day: |

# 7.1.3.2 Endpoints Other Than Fistula Assessment

All evaluable data (ie, non-missing data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day for others, the later observation will be used.

Table 7.c Visit Window of PDAI Score

| | Scheduled Stud | dy Day | Time Interval<br>(days) |
|----------|----------------|--------|-------------------------|
| Visit | (days) | | Study Day |
| Baseline | Study Day: | 1 | -39 - 1 |
| Week 2 | Study Day: | 15 | 2 - 22 |
| Week 4 | Study Day: | 29 | 23 - 43 |
| Week 8 | Study Day: | 57 | 44 - 85 |
| Week 16 | Study Day: | 113 | 86 - 141 |
| Week 24 | Study Day: | 169 | 142 - 198 |
| Week 40 | Study Day: | 281 7 | 199 - 323 |
| Week 52 | Study Day: | 365 | 324 - 448 |
| Week 104 | Study Day: | 729 | 449 - 812 |
| Week 156 | Study Day: | 1093 | 813 - |

Table 7.d Visit Window of CDAI Score

| | | Scheduled Study 1 | Dav | Time Interval<br>(days) |
|--------|----------|-------------------|------|-------------------------|
| | Visit | (days) | · _ | Study Day |
| | Baseline | Study Day: | 1 | -39 - 1 |
| | Week 24 | Study Day: | 169 | 2 - 198 |
| | Week 52 | Study Day: | 365 | 199 - 448 |
| | Week 156 | Study Day: | 1093 | 449 - |
| operty | \Qx | | | |

Table 7.e Visit Window of Van Assche Score

| Darvadstrocel-3002<br>Statistical Analysis Plan | Page 15 of 53<br>2 September 2020 | | | |
|---|---|---|---|---|
| Table 7.e Visit V | Vindow of Van Assch | e Score | | |
| | Scheduled Study | Day | Time Interval<br>(days) | Terms of Use |
| Visit | (days) | _ | Study Day | 5 |
| Baseline | Study Day: | -35 | -391 | |
| Week 24 | Study Day: | 169 | 1 - 198 | <b>√</b> Ø. |
| Week 52 | Study Day: | 365 | 199 - 448 | |
| Week 156 | Study Day: | 1093 | 449 - | 30, |
| Table 7 f Visit V | Vindow of Vital Signs | | | applicable |
| Table 7.f Visit V | Vindow of Vital Signs | <u> </u> | | 7) |
| | | | Time Interval | |
| Visit | Scheduled Study<br>(days) | Day | (days) Study Day | |
| Dasalina | Ctude Down | 1 | 20.0 | |

Table 7.f Visit Window of Vital Signs

| Scheduled Stud<br>(days) Study Day: | 1<br>15<br>29<br>57<br>113<br>69<br>281<br>365 | Time Interva<br>(days) Study Day -39 -1 2 -22 23 - 43 44 - 85 86 - 141 142 - 198 199 - 323 324 - 448 |
|---|---|---|
| Study Day: | 1<br>15<br>29<br>57<br>113<br>69<br>281<br>365 | 2 22 23 - 43 44 - 85 86 - 141 142 - 198 199 - 323 |
| Study Day: | 15<br>29<br>57<br>113<br>(69<br>281<br>365 | -39 22<br>22 23 - 43<br>44 - 85<br>86 - 141<br>142 - 198<br>199 - 323 |
| Study Day: | 15<br>29<br>57<br>113<br>(69<br>281<br>365 | 2 22<br>23 - 43<br>44 - 85<br>86 - 141<br>142 - 198<br>199 - 323 |
| Study Day: | 29<br>57<br>113<br>(69<br>281<br>365 | 23 - 43<br>44 - 85<br>86 - 141<br>142 - 198<br>199 - 323 |
| Study Day: Study Day: Study Day: Study Day: Study Day: Study Day: Study Day: | 57<br>113<br>669<br>281<br>365 | 44 - 85<br>86 - 141<br>142 - 198<br>199 - 323 |
| Study Day: Study Day: Study Day: Study Day: Study Day: Study Day: | 113<br>(69<br>281<br>365 | 86 - 141<br>142 - 198<br>199 - 323 |
| Study Day:<br>Study Day:<br>Study Day:<br>Study Day; | 281<br>365 | 142 - 198<br>199 - 323 |
| Study Day:<br>Study Day:<br>Study Day; | 281 | 199 - 323 |
| Study Day:<br>Study Day: | 365 | |
| Study Day: | <u></u> | 324 - 448 |
| | | 324 - 440 |
| S: 1 DC | 547 | 449 - 638 |
| Study Day: | 729 | 639 - 812 |
| Study Day: | 911 | 813 - 1002 |
| Study Day: | 1093 | 1003 - |
| | Study Day: | midy Day: 1093 |

Visit Window of Clinical Laboratory Tests Table 7.g

| Statistical Analysis Plan | 2 September 2020 | | | |
|---|---|---|---|---|
| Гable 7.g Visit V | Vindow of Clinical L | aboratory ' | Tests | |
| Visit | Scheduled Study<br>(days) | Day | Time Interval<br>(days)<br>Study Day | applicable rems of Us |
| Baseline | Study Day: | 1 | -39 - 1 | arrive and the second |
| Week 2 | Study Day: | 15 | 2 - 22 | 76, |
| Week 4 | Study Day: | 29 | 23 - 43 | |
| Week 8 | Study Day: | 57 | 44 - 85 | 20. |
| Week 16 | Study Day: | 113 | 86 - 141 | |
| Week 24 | Study Day: | 169 | 142 - 198 | 20% |
| Week 52 | Study Day: | 365 | 199 - 448 | , O. |
| Week 104 | Study Day: | 729 | 449 - 812 | 9 |
| Week 156 | Study Day: | 1093 | 813 - 😠 | |
| | | | -0 | |

Table 7.h

| Week 156 | Study Day: | 1093 | 813 - 💢 |
|-----------|-------------------------|--------------|-------------------------|
| Table 7.h | Visit Window of Anti-do | onor Antibo | dy Test |
| | Scheduled St | udy Day | Time Interval<br>(days) |
| Visit | (days | <i>L</i> , ( | Study Day |
| Baseline | Study Day: | (y) | -39 - 1 |
| Week 2 | Study Day: | 15 | 2 - 22 |
| Week 4 | Study Day: | 29 | 23 - 43 |
| Week 8 | Study Day; | 57 | 44 - 85 |
| Week 16 | Study Day: | 113 | 86 - 141 |
| Week 24 | Study Day: | 169 | 142 - 198 |
| Week 52 | Study Day: | 365 | 199 - 448 |
| Week 104 | Študy Day: | 729 | 449 - 812 |
| Week 156 | Study Day: | 1093 | 813 - |

# Significance Level and Confidence Coefficient

Confidence coefficient: 90% (two-sided), 95% (two-sided).

# 7.1.5 Calculation of Combined Remission, Clinical Remission, Response

Combined Remission at Week 24(Primary endpoint)

Fistula MRI assessment at Week 24(LOCF) and fistula clinical assessment at Week 24(LOCF) will be used when combined remission at Week 24 is calculated based on the definition of section 7.1.1.

If either of the two is missing, non-remission will be imputed.

If a subject received rescue therapy which is not allowed in section 7.4 of the protocol or

medications which could affect fistula closure directly prior to visit 8(Week 24) will be handled as non-remission.

- Clinical Remission, Response at Week 24(Secondary endpoint).
   Fistula clinical assessment at Week 24(LOCF) will be used when clinical remission or response at Week 24 is calculated based on the definition of section 7.1.1.

   If fistula clinical assessment is missing, non-remission(non-response) will be imputed.
   If a subject received rescue therapy which is not allowed in section 7.4 of the protocolor medications which could affect fistula closure directly prior to visit 8(Week 24) will be handled as non-remission.
- Combined Remission at Week 52(Secondary endpoint).
   Fistula MRI assessment at Week 52(LOCF) and fistula clinical assessment at Week 52(LOCF) will be used when combined remission at Week 52 is calculated based on the definition of section 7.1.1.
   If either of the two is missing, non-remission will be imputed.
- Clinical Remission, Response at Week 52(Secondary endpoint).
   Fistula clinical assessment at Week 52(LOCF) will be used when clinical remission or response at Week 52 is calculated based on the definition of section 7.1.1.
   If fistula clinical assessment is missing, non-remission(non-response) will be imputed.
- Combined Remission at Week 104/Week 156(Additional endpoint).
   Fistula MRI assessment at Week 104(LOCF)/Week 156(LOCF) and fistula clinical assessment at Week 104(LOCF)/156(LOCF) will be used when combined remission at Week 104/Week 156 are calculated based on the definition of section 7.1.1.
   If either of the two is missing, non-remission will be imputed.
- Clinical Remission, Response at Week 104/Week 156(Additional endpoint).
   Fistula clinical assessment at Week 104(LOCF)/Week 156(LOCF) will be used when clinical remission or response at Week 104/Week 156 are calculated based on the definition of section 7.1.1.
   If fistula clinical assessment is missing, non-remission(non-response) will be imputed.
- Clinical Remission, Response for Time Point Analysis(Additional endpoint).
   Fistula clinical assessment at each analysis visit after baseline in Table 7.b other than LOCF will be used when clinical remission or response for each time point analysis is calculated based on the definition of section 7.1.1.
   If fistula clinical assessment is missing, it will be handled as missing.

# 7.1.6 Calculation of Relapse in Subjects with Clinical/Combined Remission

Relapse at Week 24 in subjects with clinical remission at previous visit.

The first clinical remission date before Day 198 will be identified. Per subject with clinical remission above, subject will be defined as relapsed if there is a fistula MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the first

clinical remission and by Day 198 based on the definition of section 7.1.1. Otherwise the subject

The combined remission date at Week 24(latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 198. the subject with combined remission above and who have at least one fistula MRI assessment of >2 are with a state of the subject. with active drainage after the combined remission date and by Day 448 based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

Relapse at Week 104 in subjects with combined remission at Week 52.

The combined remission date at Week 52(latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 448, the subject will be defined as relapsed if there is a MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the combined remission date and by Day 812 based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

Relapse at Week 156 in subjects with combined remission at Week 104.

The combined remission date at Week 104(latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 812, the subject will be defined as relapsed if there is a MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the combined remission date based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

### 7.2 **Analysis Sets**

- Intention to treat (ITT): All subjects who have enrolled into treatment period.
- Modified intention to treat (mITT): All subjects who have received the study treatment and whose primary efficacy endpoint is evaluable.
- Per protocol set (PPS): All subjects who have completed the minimum protocol-specified procedures without any major protocol deviations (ie, subjects who met the following criteria will be excluded from the PPS).
  - Subjects who did not meet inclusion criteria #3, #5, #6, or #7.
  - Subjects who met exclusion criteria #1, #2, #3, #4, #5, #6, #7, #8, #9, #10, #11, #21, #23, #24, #25, or #27.

- Subjects who have violated the rules for medications and treatments specified in section 7.3 of the protocol prior to visit 8(Week 24).
- (eins of Use Subjects who have violated the rules for rescue therapy specified in section 7.4 of the protocol prior to visit 8(Week 24).
- Subjects who received less than 24 mL of the study treatment.
- Subjects who did not have either fistula MRI assessment or fistula clinical assessment 45 days prior to or post Study Day 169.
- Safety analysis set:

All subjects who have received the study treatment.

#### 7.3 **Disposition of Subjects**

#### 7.3.1 **Study Information**

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version

WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical Methods:

(1) Study Information

Study information shown in the analysis variables section will be provided.

# 7.3.2 Screen Failures

Analysis Set:

All Subjects Who Did Not Enter the Treatment Period

Analysis Variables:

Age (years)

Gender [Male, Female]

# Analytical Methods:

# (1) Screen Failures

applicable Terms of Use Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

# 7.3.3 Subject Eligibility

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

Eligibility Status

[Eligible for Entrance into the Treatment Period, Not Eligible for Entrance into the Treatment Period

Primary Reason for Subject Not Being Eligible

[Death, Adverse Event, Screen Failure, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

# Analytical Methods:

(1) Eligibility for Entrance into the Treatment Period

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will be used as the denominator.

# Number of Subjects Who Entered the Treatment Period by Site

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Status of Entrance into the Treatment Period [Entered]

Stratum:

Site [Site numbers will be used as categories]

Analytical Methods:

(1) Number of Subjects Who Entered the Treatment Period by Site

Frequency distributions will be provided for each stratum.

# 7.3.5 Disposition of Subjects for Follow-up Period

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Study Treatment Administration Status

[Eligible but Not Treated]

Reason for Not Being Treated

cable Terms of Use [Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

Completion Status for Follow-up Period

[Completed/Ongoing, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

Analytical Methods:

(1) Disposition of Subjects

Frequency distributions will be provided. When calculating percentages for the reasons for not being treated, the total number of subjects not treated will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

(2) Completion Status for Follow-up Period

Frequency distributions will be provided for Completion Status for Follow-up Period(categories of Completed, Ongoing and Prematurely Discontinued).

# **Completion Status for Follow-up Period**

Analysis Set: 40

All Subjects Who Entered the Treatment Period

Analysis Variables:

Completion Status for Follow-up Period

[Completed/Ongoing, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

# Categories:

Duration of Study after Baseline (days)

[Min - 57, 58 - 169, 170-281, 282 - Max]

# Analytical Methods:

(1) Completion Status for Follow-up Period by Duration of Study after Baseline

Frequency distributions will be provided for each category of duration of study after baseline. ift some soppies

# 7.3.7 Disposition of Subjects for Long-Term Follow-up Period

Analysis Set:

All Subjects Who Completed the Follow-up period

Analysis Variables:

Completion Status for Long-Term Follow-up Period

[Completed/Ongoing, Prematurely Discontinued

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

# Analytical Methods:

(1) Disposition of Subjects

Frequency distributions will be provided. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

(2) Completion Status for Long-Term Follow-up Period

Frequency distributions will be provided for Completion Status for Long-Term Follow-up Period (categories of Completed, Ongoing and Prematurely Discontinued).

## 7.3.8 Completion Status for Long-Term Follow-up Period

Analysis Set:

All Subjects Who Completed the Follow-up Period

Analysis Variables:

Completion Status for Long-Term Follow-up Period

[Completed/Ongoing, Prematurely Discontinued]

Reason for Discontinuation

Phicable Terms of Use [Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

Categories:

Duration of Study after Baseline (days)

[Min - 547, 548 - 729, 730-911, 912 - Max]

Analytical Methods:

(1) Completion Status for Long-Term Follow-up Period

Frequency distributions will be provided for each category of duration of study after baseline.

# 7.3.9 Protocol Deviations and Analysis Sets

# 7.3.9.1 Protocol Deviations

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Significant Protocol Deviation

[Entry Criteria, Concomitant Medication, Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria]

Analytical Methods:

(1) Protocol Deviations

Frequency distributions will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

7.3.9.2 Analysis Sets

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Handling of Subjects

[Categories are based on the specifications in Subject Evaluability List]

# **Analysis Sets**

Intention to Treat [Included] Modified Intention to Treat [Included] Per Protocol Set [Included] Safety Analysis Set [Included]

# Analytical Methods:

- (1) Subjects Excluded from Analysis Sets
- (2) Analysis Sets

Phicable Terms of Use Frequency distributions will be provided. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

## 7.4 **Demographic and Other Baseline Characteristics**

Analysis Set:

Intention to Treat

Analysis Variables:

Age (years)

[Male, Female] Gender

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$ 

Smoking Classification [Never, Current, Former]

Previous use of Antibiotics [Yes, No]

Previous use of Immunosuppressants [Yes, No]

Previous use of Biologics [Yes, No]

**Concomitant Medications** [Biologics only, Immunosuppressants only,

Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

Duration of Crohn's Disease (years)

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

[1 IO + 1 EO, 1 IO + 2 EOs, 1 IO + 3 EOs, 2 IOs + 1 EO, 2 IOs + 2 EOs, 2 IOs + 3 EOs]

Topography of Draining EOs at Screening

[0 EO, 1 EO, 2 EOs, 3EOs]

CDAI Total Score at Baseline

Analytical Methods:

(1) Summary of Demographics and Baseline Characteristics

and subject to the applica Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

## 7.5 **Medical History and Concurrent Medical Conditions**

Analysis Set:

Safety Analysis Set

Analysis Variables:

Medical History

**Concurrent Medical Conditions** 

Analytical Methods:

- (1) Medical History by System Organ Class and Preferred Term
- (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency. A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

#### 7.6 **Medication History and Concomitant Medications**

Concomitant medications whose start date occurred on or before Week 24 visit, i.e. the latest fistula clinical assessment or the latest visit by Day 198, will be summarized.

Analysis Set:

Safety Analysis Set

Analysis Variables:

**Medication History** 

**Concomitant Medications** 

- (3) Concomitant Medications That Started After Baseline by Preferred Medication Name

  (4) Concomitant Medications That Started After Baseline by Preferred Medications That Started After Baseline by Preferred Medications That Started After Baseline by Preferred Those That Concomitant Medications That Conco Those That Started After Baseline by Preferred Medication Name

Frequency distributions will be provided. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several and subject only and subject of the medications with the same preferred medication name will be counted only once for that preferred medication name.

#### 7.7 **Study Drug Exposure and Compliance**

Analysis Set:

Safety Analysis Set

Analysis Variables:

Total Exposure (mL)

Total Exposure per IOs (mL)

Total Exposure per EOs (mL)

Duration of follow-up after baseline by Week 24 (weeks)

Analytical Methods:

(1) Summary of Total Exposure

Descriptive statistics will be provided.

#### 7.8 **Efficacy Analysis**

The intention to treat will be the main analysis set used. The modified intention to treat and the per protocol set will be used for the primary and secondary endpoints in order to examine the robustness of the results.

## **Primary Endpoint** 7.8.1

# 7.8.1.1 Proportion of Subjects with Combined Remission at Week 24

# Analysis Set:

Intention to Treat

Modified Intention to Treat

Per Protocol Set

# Analysis Variables:

Combined Remission at Week 24

# Analytical Methods:

(1) Primary Analysis

two-Frequency distributions will be provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method) for the intention to treat.

(2) Secondary Analysis

Frequency distributions will be provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method) for the modified intention to treat and the per protocol set.

# **Secondary Endpoints**

Efficacy analysis using data up to Wee

# 7.8.2.1 Proportion of Subjects with Clinical Remission and Response at Week 24

# Analysis Set:

Intention to Treat

Modified Intention to Treat

Per Protocol Set

Analysis Variables:

Clinical Remission at Week 24

Response at Week 24

# Analytical Methods:

The same analysis for the primary endpoint will be performed.

# 7.8.2.2 Proportion of Subjects with Relapse at Week 24

Analysis Set:

Intention to Treat

Analysis Variables:

Relapse at Week 24

Analytical Methods:

icable Terms of Use (1) Number and Percentage of Subjects with Relapse at Week 24 Within the subjects with clinical remission at previous visit, frequency distributions will be e interest to the provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method).

# 7.8.2.3 Time to Clinical Remission and Response by Week 24

Analysis Set:

Intention to Treat

Analysis Variables:

Time to Clinical Remission by Week 24

Time to Response by Week 24

Analytical Methods:

For the following time to event analyses, subjects without event will be handled as censor at the date of last fistula clinical assessment.

- (1) Summary of Time to Event by Week 24 Frequency distribution of subjects who experienced event and who were censored will be provided. Quartiles of time to event will be estimated using the Kaplan-Meier method.
- (2) Kaplan-Meier Plot Kaplan Meier plot of time to clinical remission/response by Week 24 will be provided.

# Time to Relapse by Week 24

Analysis Set:

Intention to Treat

Analysis Variables:

Time to Relapse by Week 24

# Analytical Methods:

Within the subjects with clinical remission at previous visit, the following analyses will be performed. For the following time to event analyses, subjects without event will be handled as censor at the date of last fistula clinical assessment or last fistula MRI assessment.

- (1) Summary of Time to Event by Week 24 Frequency distribution of subjects who experienced event and who were censored will be provided. Quartiles of time to event will be estimated using the Kaplan-Meier method.
- (2) Kaplan-Meier Plot Kaplan-Meier plot of time to relapse by Week 24 will be provided.

# 7.8.2.5 PDAI Score

Analysis Set:

Intention to Treat

Analysis Variables:

PDAI Total Score

PDAI Domain Scores(Discharge, Pain/restriction of activities, Restriction of Sexual Activity, Type of Perianal Disease, Degree of Induration)

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24

Analytical Methods:

- (1) Summary of PDAI Scores and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline for each visit will be provided.
- (2) Mean and Standard Deviation Plots Mean observed values and changes from baseline will be plotted for each visit with standard deviation bars.

7.8.2.6 *CDAI Score* 

Analysis Set:

Intention to Treat

Intention to Ti
Analysis Variables:
CDAIT

**CDAI Total Score** [Min<= - <150, 150<= - <=220, 220< - <=450, 450< - <=Max]

CDAI Sub Scores

Visit:

Analytical Methods:

- Summary of CDAI Scores and Change from Baseline by Visit
  Frequency distribution for categorical variables and descriptive statistics of observed values and changes from baseline for each visit will be provided.

  Mean and Standard Deviation Plots
  Mean observed values and changes from <sup>L</sup>
  deviation bars. (1) Summary of CDAI Scores and Change from Baseline by Visit
- (2) Mean and Standard Deviation Plots use only and subject to the app

# 7.8.2.7 Van Assche Score

Analysis Set:

Intention to Treat

Analysis Variables:

Van Assche Total Score

Van Assche Domain Scores

Visit:

Baseline, Week 24

Analytical Methods:

- (1) Summary of Van Assche Scores and Change from Baseline by Visit Frequency distribution for categorical variables and descriptive statistics of observed values and changes from baseline for each visit for continuous variables will be provided.
- (2) Mean and Standard Deviation Plots Mean observed values and changes from baseline will be plotted for each visit with standard deviation bars for continuous variables.

# **Additional Endpoints**

Efficacy analysis using data up to Week 24

7.8.3.1 Timepoint Analysis of Clinical Remission and Response

Analysis Set:

Intention to Treat

Analysis Variables:

Clinical Remission

Response

Visit:

Week 2, Week 4, Week 8, Week 16, Week 24

Analytical Methods:

The same analysis for the primary endpoint will be performed by visit.

# Statistical/Analytical Issues

7.8.4.1 Adjustments for Covariates

Not applicable.

# 7.8.4.2 Handling of Dropouts or Missing Data

applicable reims of Use Values below the lower limit of quantification will be treated as zero when calculating the descriptive statistics. Values above the upper limit of quantification will be treated as the upper limit of quantification when calculating the descriptive statistics.

For combined remission, clinical remission, response

For the primary and secondary analyses of the primary endpoint, the last observation carried forward (LOCF) from the latest earlier post-baseline visit (including an Early Termination Visit prior to Week 24, if applicable) will apply in case of missing clinical assessment at Week 24. In case of missing MRI data at Week 24, LOCF from an Early Termination Visit prior to Week 24 will apply if applicable. In case of no MRI data by Week 24 or no post-baseline clinical assessment, non-response will be imputed. If rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly occur prior to visit 8(Week 24), non-response will be imputed overriding all other imputation conventions.

The handling above for the primary endpoint will also be applied to proportion of subjects with clinical remission at Week 24, proportion of subjects with response at Week 24 and proportion of subjects with combined remission at Week 52.

# 7.8.4.3 Multicenter Studies

Although this study is a multicenter study, treatment-by-center interaction will not be explored since the number of subjects for each center is not sufficient for such exploration.

7.8.4.4 Multiple Comparison/Multiplicity

Not applicable.

# 7.8.4.5 Use of an "Efficacy Subset" of Subjects

In addition to analyses on the primary endpoint using the intention to treat, a secondary analysis will also be performed using the modified intention to treat and the per protocol set to confirm the robustness of the results.

# only and subject to the applicable Terms of Use 7.8.4.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

Not applicable.

# 7.8.4.7 Examination of Subgroups

# Efficacy analysis using data up to Week 24

Analysis Set:

Intention to treat

Analysis Variables:

Combined Remission at Week 24

Clinical Remission at Week 24

Response at Week 24

Subgroups:

Age 
$$[Min \le - \le 65, 65 \le - \le Max]$$

Gender [Male, Female]

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

$$[1 \text{ IO} + 1 \text{ EO}, 1 \text{ IO} + (2 \le \text{EOs}), 2 \text{ IOs} + (1 \le \text{EOs})]$$

Previous use of Antibiotics

[Yes, No]

Previous use of Immunosuppressants [Yes, No]

Previous use of Biologics [Yes, No]

**Concomitant Medications** [Biologics only, Immunosuppressants only, Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

Analytical Methods:

# (1) Descriptive Statistics

Frequency distributions will be provided for above each subgroups.

# **Other Outcomes**

Not applicable.

#### 7.10 **Safety Analysis**

Safety analysis using data up to Week 24

# 7.10.1 Adverse Events

t [Related, Not Related]
[Mild, Moderate, Severe]

provided.
tverse Events

Events TEAEs whose date of onset occurred on or before Week 24 visit, i.e. the latest fistula clinical assessment or the latest visit by Day 198, will be summarized.

7.10.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

Categories:

Relationship to Study Treatment [Related, Not Related]

Intensity

Analytical Methods:

The following summaries will be provided.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 2) Relationship of Treatment-Emergent Adverse Events to study treatment (number of events, number and percentage of subjects).
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 4) Treatment-Emergent Adverse Events leading to study discontinuation (number of events, number and percentage of subjects).
  - 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 6) Relationship of serious Treatment-Emergent Adverse Events to study treatment (number of events, number and percentage of subjects).
  - 7) Serious Treatment-Emergent Adverse Events leading to study discontinuation (number of events, number and percentage of subjects).
  - Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects).

TEAEs will be counted according to the rules below.

# Number of subjects

Summaries for 2) and 6)

A subject with occurrences of TEAE in both categories (ie, Related and Not Related) will be counted once in the Related category.

Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

Summaries other than 2), 3), and 6)

A subject with multiple occurrences of TEAE will be counted only once

# Number of events

For each summary, the total number of events will be calculated. .181 subject and subject see only and subject see

7.10.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variables:

TEAE

Categories:

[Mild, Moderate, Severe] Intensity

- 57, 58 - 169, 170-281, 282 - Max] Time of Onset (day)

Analytical Methods:

The following summaries will be provided using frequency distribution.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Study Treatment-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (6) Intensity of Study Treatment-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (10) Treatment-Emergent Adverse Events of Special Interest by System Organ Class and Preferred Term
- (11) Product Malfunction-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distributions will be provided according to the rules below.

# Number of subjects

• Summary tables other than (5), (6) and (9)

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.

• Summary tables for (5) and (6)

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.

• Summary table for (9)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. Percentages will be based on the number of subjects in the safety analysis set.

7.10.1.3 Subgroup Analysis of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE**
## Subgroups:

 $[Min \le - \le 65, 65 \le - \le Max]$ Age

Gender [Male, Female]

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

 $[1 EO, 2 \leq EOs]$ 

Previous use of Antibiotics [Yes, No]

Previous use of Immunosuppressants [Yes, No]

Previous use of Biologics [Yes, No]

to the applicable remes of Use [Biologics only, Immunosuppressants only, **Concomitant Medications** 

Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

## Analytical Methods:

The following summaries will be provided for each subgroup using frequency distribution. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT.

(1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set for each subgroup.

## 7.10.1.4 Displays of Pretreatment Events

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

PTE

# Analytical Methods:

The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term.
- (2) Serious Pretreatment Events by System Organ Class and Preferred Term.

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

2 Clinical Laboratory Evaluations

2.1 Hematology and Serum Chemistry

ysis Set:

Safety Analysis Set

rsis Variables:

Hematology

Hemoglobin, Hematocrit, Red blood cells count Mean Corpuscular Hemoglobin and

## 7.10.2 Clinical Laboratory Evaluations

7.10.2.1 Hematology and Serum Chemistry

Analysis Set:

Analysis Variables:

Mean Corpuscular Hemoglobin, Mean Corpuscular Hemoglobin Concentration, White blood cells count, differential WBC (Neutrophils, Basophils, Eosinophils, Lymphocytes, Monocytes), Platelet count

Serum Chemistry

C-reactive protein, ALT, AST, Alkaline phosphatase, Gamma-glutamyl transpeptidase, Total bilirubin, Total protein, Glucose, Creatinine, Creatine phosphokinase, Blood urea nitrogen, Potassium, Sodium, Chloride

Visit:

Baseline, Week 2, Week 4 Week 8, Week 16, Week 24

Analytical Methods:

For each variable, summaries (1) to (3) will be provided.

(1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Summary of Shifts of Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

For each laboratory test, the laboratory values will be classified as "Low", "Normal"

and subject to the applicable Terms of Use or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

## 7.10.2.2 *Urinalysis*

## Analysis Set:

Safety Analysis Set

## Analysis Variables:

Specific Gravity

pН

[-, +-, +, 2+, 3+]Glucose

Protein [-, +-, +, 2+, 3+]

[-, +, 2+, 3+]Occult blood

[-, +-, +, 2+, 3+]Ketone body

[-, +, 2+, 3+]Bilirubin

[+-, +, 2+, 3+]Urobilinogen

## Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24

## Analytical Methods:

For specific gravity, summaries (1), (2) and (4) will be provided.

For pH, summary (4) will be provided.

For each variable other than specific gravity or pH, summaries (3) and (4) will be provided.

(1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Number of Subjects in Categories of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

(4) Summary of Shifts of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

Late

Lood Pressure

Lat Rate

it:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24 Live vical Methods:

For each variable, summaries (1) and (2) will be pro

) Summary of Vital Signs Parameters and Descriptive statistics for obouill be provided.

Case Plots

Plots

## 7.10.3 Vital Signs

Analysis Set:

Analysis Variables:

Visit:

Analytical Methods:

Plots over time for each subject will be presented.

# 7.10.4 Other Observations Related to Safety

7.10.4.1 Donor Specific Antibody

Analysis Set:

Safety Analysis Set

Analysis Variables:

Donor Specific Antibody

[Presence, Absence]

(Categories used in analytical methods (1) and (2))

[Presence at baseline and Presence during post-baseline, Presence at baseline and Absence during post-baseline, Absence at baseline and Presence during post-baseline,

Absence at baseline and Absence during post-baseline] (Categories used in analytical methods (3) and (4))

[Presence during post-baseline, Absence during post-baseline] (Categories used in analytical method (4))

(Presence/Absence at baseline is results of anti-HLA antibody.)

(Presence/Absence during post-baseline is results of donor specific antibody during post-baseline by Week 24, i.e. Presence if any positive results during post-baseline by Week 24, Absence if no positive results during post-baseline by Week 24.)

## Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24

## Analytical Methods:

(1) Summary of Donor Specific Antibody by Visit

Frequency distributions for each visit will be provided.

(2) Summary of Shifts of Donor Specific Antibody

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

(3) Number of Subjects in Categories of Donor Specific Antibody

Frequency distributions of results at baseline and during post-baseline will be provided.

(4) Subgroup Analysis of Efficacy and Safety Endpoints by Donor Specific Antibody

The same analyses of Section 7.8.4.7 and 7.10.1.3 will be conducted for each subgroup of Donor Specific Antibody.

7.10.4.2 Displays of Treatment-Emergent Adverse Events (Japanese)

## Analysis Set:

Safety Analysis Set

Analysis Variables:

TEAE

## Analytical Methods:

TEAEs will be summarized in the same way as in section 7.10.1.2 and 7.10.1.3. All summaries will be presented in Japanese.

## 7.11 **Interim Analysis**

There will not be any interim analysis. Note, the analysis using data up to Week 24 is the primary analysis for marketing application. Additionally, separate analyses using data up to Week 52 and overall data will be performed after all subjects complete Week 52 and Week 156 respectively.

## 7.12 **Changes in the Statistical Analysis Plan**

The analyses in the statistical analysis plan do not differ from the analyses specified in the ine appli protocol.

Changes from the previous version are listed below.

Page 11, Section 7.1.1

**Existing Text** 

(new)

Response: Defined as the clinically confirmed closure of at least 50% of all treated external openings that were draining at the screening despite gentle finger compression.

## Revised Text

- Duration of follow-up after baseline by Week 24 (weeks): (Date of the latest fistula clinical assessment or the latest visit by Day 198 – date of study treatment administration + 1)/7.
- Response: Defined as the clinically confirmed closure of at least 50% of all treated external openings that were draining at the screening despite gentle finger compression. Note: Clinically confirmed closure of at least 50% is defined as 1 closure for subjects with 1 baseline external opening, 1 or 2 closures for subjects with 2 baseline external openings, and 2 or 3 closures for subjects with 3 baseline external openings.

Rationale for Amendment

Added the definition of duration of follow-up after baseline by Week 24 and clarification of the definition of clinically confirmed closure of at least 50% in each case.

Page 12, Section 7.1.1

Existing Text

(new)

Revised Text

Presence/Absence of donor specific antibody: Results for each post-baseline visit will be presence when at least one of donor specific antibody tests (Class I and/or Class II) is presence, otherwise results will be absence. A result at baseline will represent presence/absence of anti-HLA Class I and Class II antibody.

| | nai score. CD<br>oe treated as - | AI total score and body v<br>10. | weight will be | Cut-011 by -10 | , i.e. score below - |
|---|---|---|---|---|---|
| Rationale for | r Amendmen | t | | | |
| Clarification<br>of CDAI sco | of the defini | tion of Presence/Absence | e of donor spec | cific antibody | and to add cut-off |
| Page 13, Sec | etion 7 1 3 1 | | | | able |
| Existing Tex | | | | | dico |
| Table 7.i | | low of Fistula MRI Asses | ssment | | 364 |
| 14010 / 11 | 1220 11 111 | Time Interval (days) | | sy's | |
| Vi | isit | Study Day | | ×0 | |
| Bas | seline | <u>-39</u> - Day Before<br>Preparation | | ect | |
| Wee | ek 24 | 1 - 198 | | )> | |
| Wee | ek 52 | 199 - 448 | 2 | | |
| | k 104 | 449 - 812 | aille | | |
| | k 156 | 813 - | H | | |
| | 4(LOCF) | 1 - 198 | | | |
| | 2(LOCF) | 1 - 448 | | | |
| | 04(LOCF) | 1 - 812 | | | |
| Week 15 | 56(LOCF) | 1-0 | | | |
| Table 7.j | Visit Wind | low of Fistula Clinical A | ssessment | | |

| Darvadstrocel-3002<br>Statistical Analysis Plan | | Page 43 of 53<br>2 September 2020 |
|---|---|---|
| | Time Interval (days) | · C. |
| Visit | Study Day | , 13 |
| Baseline | <u>-39</u> - Day Before<br>Preparation | 2 September 2020 2 September 2020 2 September 2020 3 September 2020 |
| Week 2 | 1 - 22 | ille |
| Week 4 | 23 - 43 | é, |
| Week 8 | 44 - 85 | |
| Week 16 | 86 - 141 | |
| Week 24 | 142 - 198 | i,Co |
| Week 40 | 199 - 323 | 00 |
| Week 52 | 324 - 448 | OX. |
| Week 104 | 449 - 812 | *//6 |
| Week 156 | 813 - | *O |
| Week 2(LOCF) | 1 - 22 | |
| Week 4(LOCF) | 1 - 43 | |
| Week 8(LOCF) | 1 - 85 | |
| Week 16(LOCF) | 1 - 141 | A S |
| Week 24(LOCF) | 1 - 198 | are |
| Week 40(LOCF) | 1 - 323 | H |
| Week 52(LOCF) | 1 - 448 | |
| Week 104(LOCF) | 1 - 812 | <i>'</i> |
| Week 156(LOCF) | 1- 15 | |

Revised Text

Visit Window of Fistula MRI Assessment Table 7.k

| | <u>Scheduled</u> | Study Day | Time Interval (days) |
|---|---|---|---|
| Visit | <u>(da</u> | <u>ys)</u> | Study Day |
| Baseline | Study Day: | Day Before<br>Preparation | - Day Before Preparation |
| Week 24 | Study Day: | <u>169</u> | <u>2</u> – 198 |
| Week 52 | Study Day: | <u>365</u> | 199 – 448 |
| Week 104 | Study Day: | 729 | 449 – 812 |
| Week 156 | Study Day: | 1093 | 813 - |
| Week 24(LOCF) | Study Day: | | <u>2</u> - 198 |
| Week 52(LOCF) | Study Day: | | <u>2</u> - 448 |
| Week 104(LOCF) | Study Day: | | <u>2</u> - 812 |
| Week 156(LOCF) | Study Day: | | <u>2</u> - |

Table 7.1 Visit Window of Fistula Clinical Assessment

| | Scheduled S | Study Day | Time Interval (days) |
|---|---|---|---|
| Visit | (day | <u>vs)</u> | Study Day |
| Baseline | Study Day: | Day Before<br>Preparation | - Day Before Preparation |
| Week 2 | Study Day: | <u>15</u> | <u>2</u> – 22 |
| Week 4 | Study Day: | <u>29</u> | 23 - 43 |
| Week 8 | Study Day: | <u>57</u> | 44 - 85 |
| Week 16 | Study Day: | <u>113</u> | 86 - 141 |
| Week 24 | Study Day: | <u>169</u> | 142 - 198 |
| Week 40 | Study Day: | <u>281</u> | 199 - 323 |
| Week 52 | Study Day: | <u>365</u> | 324 448 |
| Week 104 | Study Day: | 729 | 449 - 812 |
| Week 156 | Study Day: | 1093 | 813 - |
| Week 2(LOCF) | Study Day: | | <u>2</u> – 22 |
| Week 4(LOCF) | Study Day: | | <u>2</u> – 43 |
| Week 8(LOCF) | Study Day: | | <u>2</u> – 85 |
| Week 16(LOCF) | Study Day: | . ( | <u>2</u> – 141 |
| Week 24(LOCF) | Study Day: | RIG | <u>2</u> – 198 |
| Week 40(LOCF) | Study Day: | 0 | <u>2</u> – 323 |
| Week 52(LOCF) | Study Day: | 50 | <u>2</u> – 448 |
| Week 104(LOCF) | Study Day: | 7 | <u>2</u> – 812 |
| Week 156(LOCF) | Study Day: | | <u>2</u> - |

## Rationale for Amendment

To address scheduled study day of visit window for fistula assessment as well as other endpoints. Lower limit of time interval of baseline was removed to include all screening assessment. A subject performed fistula clinical assessment on Day 1 prior to study treatment administration. Modification to exclude Day 1 assessment prior to study treatment administration from post-baseline.

# Page 17, Section 7.1.5

# **Existing Text**

If a subject received rescue therapy which is not allowed in section 7.4 of the protocol prior to visit 8(Week 24) will be handled as non-remission.

Revised Text

... in be handled

... is be handled

... is be handled

... is a line (days)

... o - 169, 170-281, 282 - Max]

n of Study after Baseline (days)

[Min - 57, 58 - 169, 170-281, 282 - Max]

mendment

7.4

of Immunosumessa
'Internation If a subject received rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly prior to visit 8(Week 24) will be handled as non-remission.

Rationale for Amendment

To align with revised text in the protocol amendment 3 section 13.1.3.3.

## Page 22, Section 7.3.6

**Existing Text** 

Duration of Study after Baseline (days)

Revised Text

Duration of Study after Baseline (days)

Rationale for Amendment

To correct typo.

## Page 24, Section 7.4

**Existing Text** 

Previous use of Immunosupressants

Topography of Internal IOs and EOs at Baseline

[1 IO, 2 IOs]

[2 EOs, 3 EOs]

[1 IO + 2 EOs, 1 IO + 3 EOs, 2IOs + 2 EOs, 2IOs + 3 EOs]

Revised Text

Previous use of Immunosuppressants [Yes, No]

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

[1 IO + 1 EO, 1 IO + 2 EOs, 1 IO + 3 EOs, 2 IOs + 1 EO, 2 IOs + 2 EOs, 2 IOs + 3 EOs]

Concomitant medications whose start date occurred on or before Week 24 visit, i.e. the latest fistula clinical assessment or the latest visit by Day 198, will be summarized.

Rationale for Amendment

Clarification of targeted concomitant medications analyzed using 
age 26, Section 7.7

visting Text

nalveie \*\*

cialuse only and subil

Analysis Variables:

(new)

Revised Text

Analysis Variables:

Duration of follow-up after baseline by Week 24 (weeks)

Rationale for Amendment

To add summary of duration of follow-up after baseline by Week 24.


**Existing Text** 

Within the subjects with clinical remission at previous visit, the following analyses will be performed. For the following time to event analyses, subjects without event will be handled as censor at the date of last fistula clinical assessment.

Revised Text

Within the subjects with clinical remission at previous visit, the following analyses will be performed. For the following time to event analyses, subjects without event will be handled as censor at the date of last fistula clinical assessment or last fistula MRI assessment.

Rationale for Amendment

To correct appropriate text.


**Existing Text** 

In case of no MRI data by Week 24 or no post-baseline clinical assessment, non-response will be imputed. If rescue therapy which is not allowed in section 7.4 of the protocol occur prior to visit 8(Week 24), non-response will be imputed overriding all other imputation conventions.

**Revised Text** 

In case of no MRI data by Week 24 or no post-baseline clinical assessment, non-response will be imputed. If rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly occur prior to visit 8(Week 24), non-response will be imputed overriding all other imputation conventions.

Rationale for Amendment

ialuse only ar To align with revised text in the protocol amendment 3 section 13.1.3.3.


**Existing Text** 

Analysis Variables:

Combined Remission at Week 24

Subgroups:

Previous use of Immunosupressants [Yes, No]

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[2 EOs, 3 EOs]

Revised Text

Analysis Variables:

Combined Remission at Week 24

Clinical Remission at Week 24

Response at Week 24

Subgroups:

Previous use of Immunosuppressants [Yes, No]

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

 $[1 \text{ IO} + 1 \text{ EO}, 1 \text{ IO} + (2 \le \text{EOs}), 2 \text{ IOs} + (1 \le \text{EOs})]$ 

Rationale for Amendment

reins of Use of supplication the application of supplication of supplicatio To add analysis variables and subgroup category, and to correct typo and category of subgroups in topography of EOs at Baseline.

## Page 32, Section 7.10.1

**Existing Text** 

(new)

Revised Text

TEAEs whose date of onset occurred on or before Week 24 visit, i.e. the latest fistula clinical assessment or the latest visit by Day 198, will be summarized.

Rationale for Amendment

Clarification of targeted TEAEs analyzed using data up to Week 24.


**Existing Text** 

Displays of Treatment-Emergent Adverse events

**Revised Text** 

Displays of Treatment-Emergent Adverse Events

Rationale for Amendment

Property of Lake To correct typo.

Revised Text
7.10.1.3 Subgroup Analysis of Treatment-Emergent Adverse Events
Rationale for Amendment
To add subgroup analysis of TEAEs.

ge 39. Section 7.10.3
sting Text
Pulse Rate
sed Text
Leart Rate
al-

Heart Rate

Rationale for Amendment

To correct typo.

# Page 39-40, Section 7.10.4.1

**Existing Text** 

Analysis Variables:

Anti-donor Antibody [Presence, Absence]

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24

Analytical Methods:

Frequency distributions will be provided.

Revised Text

Analysis Variables:

Donor Specific Antibody

[Presence, Absence]
(Categories used in analytical methods (1) and (2))
[Presence at baseline and Presence during poor.

Presence at baseline and Absence during Absence at baseline and Presence at baseline at baseline at baseline at baseline at b

[Presence during post-baseline, Absence during post-baseline] (Categories used in analytical method (4))

(Presence/Absence at baseline is results of anti-HLA antibody.)

(Presence/Absence during post-baseline is results of donor specific antibody during postbaseline by Week 24, i.e. Presence if any positive results during post-baseline by Week 24, Absence if no positive results during post-baseline by Week 24.)

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24

Analytical Methods:

(5) Summary of Donor Specific Antibody by Visit

Frequency distributions for each visit will be provided.

(6) Summary of Shifts of Donor Specific Antibody

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

(7) Number of Subjects in Categories of Donor Specific Antibody

Frequency distributions of results at baseline and during post-baseline will be provided.

(8) Subgroup Analysis of Efficacy and Safety Endpoints by Donor Specific Antibody

The same analyses of Section 7.8.4.7 and 7.10.1.3 will be conducted for each subgroup of Donor Specific Antibody.

Existing Text

TEAEs will be summarized in the same way as in section 7.10.1.2. All summaries will be presented in Japanese.

Revised Text

TEAEs will be summarized in the same way as in section 7.10.1.2. All summaries will be presented in Japanese.

Rationale for Amendman. Proparty of Takeda. For non-commercial use only and subject to

Properly of Takeda. For non-confine cial use only and subject to the applicable Tames of Use

Properly of Takeda. For non-confine cial use only and subject to the applicable Tames of Use

# ELECTRONIC SIGNATURES

| | | ELECTRONIC SIGNATURES | 10th |
|---|---|---|---|
| | Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH:mm 'UTC') |
| Property | akeda. For hon. con | Meaning of Signature Biostatistics Approval | (dd-MMM-yyyy HH;mm 'UTC') 16-Sep-2020 02:07 UTC |



## STATISTICAL ANALYSIS PLAN

[Analysis using Data up to Week 52]

the applicable rems of Use STUDY NUMBER: Darvadstrocel-3002

A Phase 3, Multicenter, Open-Label, Uncontrolled Study to Exaliate the Efficacy and Safety of Cx601 in the Treatment of Complex Perianal Fistulas in Adult Patients with Crohn's Disease

Prepared by:

Based on:

Version: 2nd
Date: 05 March 2021 Protocol Version: Amendment 4 Protocol Date: 6 October 2020

Properly of Takeda: For non-commercial use only and subject to the applicable Terms of use

7.3.9

## TITLE PAGE Approval Signatures TABLE OF CONTENTS..... 2.0 1.0 TABLE OF CONTENTS 3 LIST OF ABBREVIATIONS 1.1 2.0 3.0 4.0 4.1 4.2 4.3 4.4 ANALYSIS ENDPOINTS......8 5.0 Primary Endpoint. 8 Secondary Endpoints 9 5.1 5.2 Safety Endpoints 9 Additional Endpoints 10 5.3 5.4 6.0 7.0 General Principles 10 7.1 Study Definitions 10 7.1.1 7.1.2 7 1 3 Definition of Study Visit Windows 12 7.1.4 7.1.5 7.1.6 7.2 7.3 Study Information 19 Screen Failures 19 7.3.3 7.3.4 Number of Subjects Who Entered the Treatment Period by Site......20 7.3.5 7.3.6 7.3.7 7.3.8

LIST OF IN-TEXT FIGURES

Figure 4.a

## 3.0 LIST OF ABBREVIATIONS

AΕ adverse event

ALP alkaline phosphatase **ALT** alanine aminotransferase AST aspartate aminotransferase **CDAI** Crohn's Disease Activity Index **DMEM** Dulbecco Modified Eagle's Medium

eASC expanded allogeneic adipose-derived stem cells

**ECG** electrocardiogram

eCRF electronic case report form **EMA** European Medicines Agency

EO **External Opening** 

Food and Drug Administration **FDA** 

**GCP** Good Clinical Practice

gamma-glutamyl transpeptidase **GGT** hepatitis B virus surface antigen HBsAg

**HBV** hepatitis B virus

hCG human chorionic gonadotropin **HCV** hepatitis C virus **HSA** human serum albumin

International Conference on Harmonisation **ICH** 

IL interleukin

interleukin international normalized ratio **INR** 

Internal Opening IO

**IRB** institutional review board

ITT intention to treat

**LOCF** last observation carried forward

MedDRA Medical Dictionary for Regulatory Activities **MHLW** Ministry of Health, Labour and Welfare

**MHRA** Medicines and Healthcare products Regulatory Agency

mITT modified intention to treat MRI magnetic resonance imaging **PCR** polymerase chain reaction **PDAI** Perianal Disease Activity Index

**PMDA** Pharmaceuticals and Medical Devices Agency

per protocol set PTE Pretreatment event SAE serious adverse event SAP statistical analysis plan

**SUSAR** suspected unexpected serious adverse reaction

| TEAE | treatment-emergent AE |
|------|-----------------------|
| TNF | tumor necrosis factor |
| ULN | upper limit of normal |
| WRC | white blood cell |

Probety of Takeda: For non-commercial life only and subject to the applicable Temps of the

## 4.0

## 4.1

To evaluate the efficacy of Cx601 for the treatment of complex perianal fistulas in adult patients with Crohn's disease over 24 weeks.

Secondary Objectives

To evaluate the efficacy of Cx601 for the treatment of complex perianal fistulas in adult patients with Crohn's disease over 24 weeks.

## 4.2

- patients with Crohn's disease over 52 weeks.
- To evaluate the safety of Cx601 for the treatment of perianal fistulas in adult patients with Crohn's disease over minimum 156 weeks.

## 4.3 **Additional Objectives**

- To evaluate the absence of clinically relevant alloreactivity
- To evaluate the effects of Cx601 on Crohn's disease activity and quality of life.

## 4.4 **Study Design**

This is Phase 3, a multicenter, open-label, uncontrolled study to evaluate the efficacy and safety of Cx601 in the treatment of complex perianal fistulas in adult patients with Crohn's disease.

Subjects with Crohn's disease whose complex perianal fistulas were previously treated and refractory (inadequate response, loss of response or intolerance) to at least one of the following treatments: antibiotics, immunosuppressants or biologics (anti-TNFs, anti-integrin or anti-IL-12/23) will be included in the study. Note that those subjects who are refractory to antibiotics only will be must be less than 25% of all subjects enrolled.

The study will permit continuation of baseline treatments for Crohn's disease in an add-on design (ie, biologics, immunosuppressants, etc.) . A total of 20 subjects are planned to be enrolled, and study product, cell suspension containing 120×10<sup>6</sup> cells of eASCs, will be intralesionally injected to all participants. Since this is the first study of Cx601 in Japanese subjects, the enrollment of at least the first 3 subjects will be adjusted not to be administered the study product at the same day.

This study consists of the screening period (approximately 5 weeks prior to study product administration, including the screening visit and the preparation visit), the treatment period (the day of study product administration), the follow-up period (approximately 52 weeks after study product administration), and the long-term follow-up period (from Week 52 to Week 156 or later; for a minimum of 104 weeks). Cx601 will be administrated once on Day 1, and the efficacy and safety of Cx601 will be mainly evaluated in the subsequent 52-week follow-up period. The primary endpoint will be evaluated at Week 24. Additionally, in the long-term follow-up period after Week 52, a safety follow-up evaluation will be performed for all subjects every 26 weeks (6 months) until Week 156 or later.

In the screening period, a screening visit (Visit 1) to determine a subject's eligibility is scheduled during the period from Day -39 to the day before preparation. All the subjects eligible by the screening will receive fistula curettage and seton placement under anesthesia at the preparation visit (Visit 2: Day -21, done no later than Day -14). Seton(s) placed will be removed on the day. of study product administration (Visit 3: Day 1), just before the administration of the study. product. Appropriate training for the preparation and the administration will be implemented to standardize the procedures between study sites.

The subjects who meet all the eligibility criteria will visit the study site on Day 1, and receive fistula curettage under anesthesia and an intralesional injection of cell suspension containing 120×10<sup>6</sup> cells of eASCs (Cx601). Thereafter, in follow-up period, the subjects will visit the study site for the clinical assessments including fistula closure at Weeks 2, 4, 8, 16, 24, 40 and 52. Radiological assessments (MRI) of fistula closure will also be performed at Weeks 24 and 52.

Additionally, in the long-term follow-up period, the safety follow-up will be performed on all the subjects (where possible) every 26 weeks (6 months) from a visit in Week 52 through Week 156. This study will be switched to a post-marketing clinical study if Cx601 is approved before the study completion.

A schematic study design is shown in Figure 4.a.

Figure 4.a **Schematic Study Design** 



## ANALYSIS ENDPOINTS

## **Primary Endpoint**

Proportion of subjects with combined remission at Week 24.

## 5.2 Secondary Endpoints

## Efficacy analysis using data up to Week 24:

- Proportion of subjects with clinical remission at Week 24.
- Proportion of subjects with response at Week 24.
- Time to clinical remission by Week 24.
- Time to response by Week 24.
- Proportion of subjects with relapse at Week 24 in subjects with clinical remission at previous visit.
- Time to relapse by Week 24 in subjects with clinical remission at previous visit.
- PDAI score (including total score, discharge sub-score and pain sub-score) up to Week 24.
- CDAI score up to Week 24.
- Van Assche score up to Week 24.

## Efficacy analysis using data up to Week 52:

- Proportion of subjects with combined remission at Week 52.
- Proportion of subjects with clinical remission at Week 52.
- Proportion of subjects with response at Week 52.
- Time to combined remission by Week 52.
- Time to clinical remission by Week 52.
- Time to response by Week 52.
- Proportion of subjects with relapse at Week 52 in subjects with combined remission at Week 24.
- Time to relapse by Week 52 in subjects with combined remission at Week 24.
- PDAI score (including total score, discharge sub-score and pain sub-score) up to Week 52.
- CDAI score up to Week 52.
- Van Assche score up to Week 52.

## 5.3 Safety Endpoints

- Adverse events (AEs) including serious adverse events (SAEs) and AEs of special interest.
- Product malfunctions.
- Physical examination findings.

- Vital signs (heart rate, blood pressure, body temperature).
- Clinical laboratory test results (serum chemistry, hematology and urinalysis).

## 5.4 Additional Endpoints

• Presence/absence of anti-donor antibody.

## 6.0 DETERMINATION OF SAMPLE SIZE

The planned sample size is 20 based on feasibility. However, this study has at least 94% probability to show a proportion of subjects with combined remission of 35% or more given an expected proportion of subjects with combined remission of 50% based on Week 24 results in the Cx601-0302 study.

# 7.0 METHODS OF ANALYSIS AND PRESENTATION

## 7.1 General Principles

## 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE) An adverse event whose date of onset occurs on or after receiving study treatment.
- Pretreatment event (PTE): Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to study treatment administration.
- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles.
- Duration of study after baseline (days): Date of last visit/contact date of study treatment administration + 1.
  - If subject is ongoing, date of last visit/contact will be imputed by date of data cut off.
- Duration of follow-up after baseline by Week 52 (weeks): (Date of the latest fistula clinical assessment or the latest visit by Day 448 date of study treatment administration + 1)/7.
- Duration of Crohn's Disease (years): (Date of informed consent date of Crohn's disease diagnosis)/365.25.
  - (If month of diagnosis is missing, month will be replaced with January. If day of diagnosis is missing, day will be replaced with 1<sup>st</sup>.)
- Combined remission: Defined as the clinically confirmed closure of all treated external openings that were draining at the screening despite gentle finger compression, and absence of collections >2 cm in the treated fistulas which is confirmed by the central MRI assessment

(a collection >2 cm is considered as present if at least two out of the 3 dimensions centrally assessed are >2 cm in any of fistula tract).

- Clinical remission: Defined as the clinically confirmed closure of all treated external openings that were draining at the screening despite gentle finger compression.
- Response: Defined as the clinically confirmed closure of at least 50% of all treated external openings that were draining at the screening despite gentle finger compression. Note: Clinically confirmed closure of at least 50% is defined as 1 closure for subjects with 1 baseline external opening, 1 or 2 closures for subjects with 2 baseline external openings, and 2 or 3 closures for subjects with 3 baseline external openings.
- Relapse: Defined as the clinically confirmed reopening of any of the treated external openings with active drainage, or the development of a collection >2 cm in the treated fistulas confirmed by central MRI assessment (a collection >2 cm is considered as present if at least two out of the 3 dimensions centrally assessed are >2 cm in any of fistula tract).
- Time to combined remission/clinical remission/response (days): The time from the study treatment administration to the first visit by which combined remission/clinical remission/response is observed.
   For combined remission, date is the latest of fistula MRI assessment and fistula clinical assessment.
- Time to relapse (days): The time from the first visit which clinical remission is observed to
  the first visit by which relapse is observed.
   (Time to relapse by Week 52 in subjects who achieved combined remission at Week 24 is
  defined as "the time from the combined remission at Week 24 to the first visit by which
  relapse is observed.)
- Presence/Absence of donor specific antibody: Results for each post-baseline visit will be
  presence when at least one of donor specific antibody tests (Class I and/or Class II) is
  presence, otherwise results will be absence. A result at baseline will represent
  presence/absence of anti-HLA Class I and Class II antibody.
- CDAI total score: CDAI total score and body weight will be cut-off by -10, ie, score below 10 will be treated as -10.

## 7.1.2 Definition of Study Days

The following definitions and calculation formulas will be used.

• Study Day: The day before study treatment administration will be defined as Study Day -1 and the day of the study treatment administration will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the study treatment administration, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.

## 7.1.3 Definition of Study Visit Windows

When calculating Study Day relative to a reference date (ie, study treatment administration [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

## 7.1.3.1 Fistula Assessment

All evaluable data (ie, non-missing data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the largest Study Day will be used.

Table 7.a Visit Window of Fistula MRI Assessment

| Fisit seline Study Da eek 24 Study Da eek 52 Study Da eek 104 Study Da ek 105 Study Da ek 156 Study Da 24(LOCF) Study Da 52(LOCF) Study Da | Preparation ay: 169 ay: 365 ay: 729 ay: 1093 ay: ay: ay: | Time Interval (da<br>Study Day - Day Before Prepar 2 - 198 199 - 448 449 - 812 813 - 2 - 198 2 - 448 2 - 812 2 - 812 2 - | |
|---|---|---|---|
| seline Study Da eek 24 Study Da eek 52 Study Da eek 104 Study Da eek 156 Study Da 24(LOCF) Study Da 52(LOCF) Study Da | Day Before Preparation ay: 169 ay: 365 ay: 729 ay: 1093 ay: ay: ay: ay: | - Day Before Preparents - 198 | ration |
| eek 24 Study Da eek 52 Study Da ek 104 Study Da ek 156 Study Da 24(LOCF) Study Da 52(LOCF) Study Da | Preparation ay: 169 ay: 365 ay: 729 ay: 1093 ay: ay: ay: | 2 - 198<br>199 - 448<br>449 - 812<br>813 -<br>2 - 198<br>2 - 448<br>2 - 812 | ration |
| eek 52 Study Da ek 104 Study Da ek 156 Study Da 24(LOCF) Study Da 52(LOCF) Study Da | ay: 365<br>ay: 729<br>ay: 1093<br>ay: ay: | 199 - 448<br>449 - 812<br>813 -<br>2 - 198<br>2 - 448<br>2 - 812 | |
| ek 104 Study Da ek 156 Study Da 24(LOCF) Study Da 52(LOCF) Study Da | ay: 729<br>ay: 1093<br>ay:<br>ay: | 449 - 812<br>813 -<br>2 - 198<br>2 - 448<br>2 - 812 | |
| ek 156 Study Da<br>24(LOCF) Study Da<br>52(LOCF) Study Da | ay: 1093<br>ay:<br>ay:<br>ay: | 813 -<br>2 - 198<br>2 - 448<br>2 - 812 | |
| 24(LOCF) Study Da<br>52(LOCF) Study Da | ay:<br>ay: | 2 - 198<br>2 - 448<br>2 - 812 | |
| 52(LOCF) Study Da | ay: | 2 - 448<br>2 - 812 | |
| | ау: | 2 - 812 | |
| 04(LOCF) Study Da<br>56(LOCF) Study Da | | | |
| 56(LOCF) Study Da | ay: | 2 - | |
| 56(LOCF) Study Da | | | |

Table 7.b Visit Window of Fistula Clinical Assessment

| | Scheduled Study Day | | Time Interval (days) |
|---|---|---|---|
| Visit | (da | | Study Day |
| Baseline | Study Day: | Day Before<br>Preparation | - Day Before Preparation |
| Week 2 | Study Day: | 15 | 2 - 22 |
| Week 4 | Study Day: | 29 | 23 - 43 |
| Week 8 | Study Day: | 57 | 44 - 85 |
| Week 16 | Study Day: | 113 | 86 - 141 |
| Week 24 | Study Day: | 169 | 142 - 198 |
| Week 40 | Study Day: | 281 | 199 - 323 |
| Week 52 | Study Day: | 365 | 324 - 448 |
| Week 104 | Study Day: | 729 | 449 - 812 |
| Week 156 | Study Day: | 1093 | 813 - |
| Week 2(LOCF) | Study Day: | 29 | 2 - 22 |
| Week 4(LOCF) | Study Day: | 200 | 2 - 43 |
| Week 8(LOCF) | Study Day: | 12/0 | 2 - 85 |
| Week 16(LOCF) | Study Day: | 20/3 | 2 - 141 |
| Week 24(LOCF) | Study Day: | 0, | 2 - 198 |
| Week 40(LOCF) | Study Day: | (5) | 2 - 323 |
| Week 52(LOCF) | Study Day: | <i></i> | 2 - 448 |
| Week 104(LOCF) | Study Day: | | 2 - 812 |
| Week 156(LOCF) | Study Day: | | 2 - |

# 7.1.3.2 Endpoints Other Than Fistula Assessment

All evaluable data (ie non-missing data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day for others, the later observation will be used.

Table 7.c Visit Window of PDAI Score

| arvadstrocel-3002<br>tatistical Analysis Plan | | | | <br>05 March 2021 |
|---|---|---|---|---|
| Table 7.c Visit W | 05 March 2021 Of March 2021 Of March 2021 | | | |
| | Scheduled Study | Day | Time Interval<br>(days) | |
| Visit | (days) | | Study Day | Λ0. |
| Baseline | Study Day: | 1 | -39 - 1 | |
| Week 2 | Study Day: | 15 | 2 - 22 | |
| Week 4 | Study Day: | 29 | 23 - 43 | - |
| Week 8 | Study Day: | 57 | 44 - 85 | |
| Week 16 | Study Day: | 113 | 86 - 141 | - 02 |
| Week 24 | Study Day: | 169 | 142 - 198 | |
| Week 40 | Study Day: | 281 | 199 - 323 | ₹3° |
| Week 52 | Study Day: | 365 | 324 - 448 | - |
| Week 104 | Study Day: | 729 | 449 - 812 | - |
| Week 156 | Study Day: | 1093 | 813 - | _ |

Visit Window of CDAI Score Table 7.d

| | Scheduled Study D | ayon | Time Interval<br>(days) |
|----------|-------------------|------|-------------------------|
| Visit | (days) | | Study Day |
| Baseline | Study Day: | 1 | -39 - 1 |
| Week 24 | Study Day: O | 169 | 2 - 198 |
| Week 52 | Study Day: | 365 | 199 - 448 |
| Week 156 | Study Day: | 1093 | 449 - |

Visit Window of Van Assche Score Table 7.e

| LOT | Scheduled Study | Day | Time Interval<br>(days) |
|----------|-----------------|------|-------------------------|
| Visit | (days) | | Study Day |
| Baseline | Study Day: | -35 | -391 |
| Week 24 | Study Day: | 169 | 1 - 198 |
| Week 52 | Study Day: | 365 | 199 - 448 |
| Week 156 | Study Day: | 1093 | 449 - |

Visit Window of Vital Signs Table 7.f

| Darvadstrocel-3002<br>Statistical Analysis Plan | | | | 05 March 2021 |
|---|---|---|---|---|
| Γable 7.f Visit V | Vindow of Vital Signs | <b>.</b> | | |
| | Scheduled Study | Dov | Time Interval<br>(days) | ring . |
| Visit | (days) | Day | Study Day | 10° |
| Baseline | Study Day: | 1 | -39 - 1 | |
| Week 2 | Study Day: | 15 | 2 - 22 | |
| Week 4 | Study Day: | 29 | 23 - 43 | -<br>''C'O' |
| Week 8 | Study Day: | 57 | 44 - 85 | |
| Week 16 | Study Day: | 113 | 86 - 141 | |
| Week 24 | Study Day: | 169 | 142 - 198 | - CO |
| Week 40 | Study Day: | 281 | 199 - 323 | |
| Week 52 | Study Day: | 365 | 324 - 448 | - |
| Week 78 | Study Day: | 547 | 449 - 638 | - |
| Week 104 | Study Day: | 729 | 639 - 812 | - |
| Week 130 | Study Day: | 911 | 813 - 1002 | - |
| Week 156 | Study Day: | 1093 | 1003 - | - |

Visit Window of Clinical Laboratory Tests Table 7.g

| | Scheduled Study | Time Interval<br>(days) | |
|----------|-----------------|-------------------------|-----------|
| Visit | (days) | | Study Day |
| Baseline | Study Day: | 1 | -39 - 1 |
| Week 2 | Study Day: | 15 | 2 - 22 |
| Week 4 | Study Day: | 29 | 23 - 43 |
| Week 8 | Study Day: | 57 | 44 - 85 |
| Week 16 | Study Day: | 113 | 86 - 141 |
| Week 24 | Study Day: | 169 | 142 - 198 |
| Week 52 | Study Day: | 365 | 199 - 448 |
| Week 104 | Study Day: | 729 | 449 - 812 |
| Week 156 | Study Day: | 1093 | 813 - |

Week 156

| Darvadstrocel-3002<br>Statistical Analysis Plan | | | | <br>05 March 2021 |
|---|---|---|---|---|
| Table 7.h Visit W | indow of Anti-dono | r Antibody | y Test | 03 March 2021 |
| | Scheduled Study | Dav | Time Interval<br>(days) | applicable Terms of |
| Visit | (days) | · | Study Day | √⊗, |
| Baseline | Study Day: | 1 | -39 - 1 | |
| Week 2 | Study Day: | 15 | 2 - 22 | |
| Week 4 | Study Day: | 29 | 23 - 43 | - 11CO |
| Week 8 | Study Day: | 57 | 44 - 85 | - 10°C |
| Week 16 | Study Day: | 113 | 86 - 141 | |
| Week 24 | Study Day: | 169 | 142 - 198 | - CO |
| Week 52 | Study Day: | 365 | 199 - 448 | <b>V</b> |
| Week 104 | Study Day: | 729 | 449 - 812 | - |

Visit Window of Anti-donor Antibody Test Table 7.h

## 7.1.4 Significance Level and Confidence Coefficient

Confidence coefficient: 90% (two-sided), 95% (two-sided).

Study Day:

## Calculation of Combined Remission, Clinical Remission, Response 7.1.5

Combined Remission at Week 24(Primary endpoint)

Fistula MRI assessment at Week 24(LOCF) and fistula clinical assessment at Week 24(LOCF) will be used when combined remission at Week 24 is calculated based on the definition of section 7.1.1.

1093

If either of the two is missing, non-remission will be imputed.

If a subject received rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly prior to visit 8(Week 24) will be handled as non-remission.

- Clinical Remission, Response at Week 24(Secondary endpoint). Fistula clinical assessment at Week 24(LOCF) will be used when clinical remission or response at Week 24 is calculated based on the definition of section 7.1.1. If fistula clinical assessment is missing, non-remission(non-response) will be imputed. If a subject received rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly prior to visit 8(Week 24) will be handled as non-remission.
- Combined Remission at Week 52(Secondary endpoint). Fistula MRI assessment at Week 52(LOCF) and fistula clinical assessment at Week 52(LOCF) will be used when combined remission at Week 52 is calculated based on the definition of section 7.1.1.

If either of the two is missing, non-remission will be imputed.

- Clinical Remission, Response at Week 52(Secondary endpoint).
   Fistula clinical assessment at Week 52(LOCF) will be used when clinical remission or response at Week 52 is calculated based on the definition of section 7.1.1.
   If fistula clinical assessment is missing, non-remission(non-response) will be imputed.
- Combined Remission at Week 104/Week 156(Additional endpoint).
   Fistula MRI assessment at Week 104(LOCF)/Week 156(LOCF) and fistula clinical assessment at Week 104(LOCF)/156(LOCF) will be used when combined remission at Week 104/Week 156 are calculated based on the definition of section 7.1.1.
   If either of the two is missing, non-remission will be imputed.
- Clinical Remission, Response at Week 104/Week 156(Additional endpoint).
   Fistula clinical assessment at Week 104(LOCF)/Week 156(LOCF) will be used when clinical remission or response at Week 104/Week 156 are calculated based on the definition of section 7.1.1.

   If fistula clinical assessment is missing, non-remission(non-response) will be imputed.
- Clinical Remission, Response for Time Point Analysis(Additional endpoint).
   Fistula clinical assessment at each analysis visit after baseline in Table 7.b other than LOCF will be used when clinical remission or response for each time point analysis is calculated based on the definition of section 7.1.1.
   If fistula clinical assessment is missing, it will be handled as missing.

## 7.1.6 Calculation of Relapse in Subjects with Clinical/Combined Remission

• Relapse at Week 24 in subjects with clinical remission at previous visit.

The first clinical remission date before Day 198 will be identified. Per subject with clinical remission above, subject will be defined as relapsed if there is a fistula MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the first clinical remission and by Day 198 based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

• Relapse at Week 52 in subjects with combined remission at Week 24.

The combined remission date at Week 24(latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 198, the subject will be defined as relapsed if there is a MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the combined remission date and by Day 448 based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

• Relapse at Week 104 in subjects with combined remission at Week 52.

The combined remission date at Week 52(latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 448, the subject will be defined as relapsed if there is a MRI assessment of >2 cm or a clinical assessment of reopening of external openings
Day 812 based on the definition of Day 812 based on the definition of Day Bay 812 based on the definition of Day 812 base section 7.1.1. Otherwise the subject will be defined as non-relapsed.

#### 7.2 **Analysis Sets**

- Intention to treat (ITT): All subjects who have enrolled into treatment period.
- Modified intention to treat (mITT): All subjects who have received the study treatment and whose primary efficacy endpoint is evaluable.
- Per protocol set (PPS):

All subjects who have completed the minimum protocol-specified procedures without any major protocol deviations (ie, subjects who met the following criteria will be excluded from the PPS).

- Subjects who did not meet inclusion criteria #3, #5, #6, or #7.
- Subjects who met exclusion criteria #1, #2, #3, #4, #5, #6, #7, #8, #9, #10, #11, #21, #23, #24, #25, or #27.
- Subjects who have violated the rules for medications and treatments specified in section 7.3 of the protocol prior to visit 8 (Week 24).
- Subjects who have violated the rules for rescue therapy specified in section 7.4 of the protocol prior to visit 8 (Week 24).
- Subjects who received less than 24 mL of the study treatment.
- Subjects who did not have either fistula MRI assessment or fistula clinical assessment 45 days prior to or post Study Day 169.
- Safety analysis set:

All subjects who have received the study treatment.

## 7.3 Disposition of Subjects

#### 7.3.1 Study Information

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version

WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical Methods:

(1) Study Information

Study information shown in the analysis variables section will be provided.

#### 7.3.2 Screen Failures

Analysis Set:

All Subjects Who Did Not Enter the Treatment Period

Analysis Variables:

Age (years)

Gender [Male, Female]

Analytical Methods

(1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

# 7.3.3 Subject Eligibility

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

Eligibility Status

[Eligible for Entrance into the Treatment Period, Not Eligible for Entrance into the Treatment Period]

Primary Reason for Subject Not Being Eligible

reins of Use [Death, Adverse Event, Screen Failure, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

## Analytical Methods:

(1) Eligibility for Entrance into the Treatment Period

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will be used as the denominator.

#### Number of Subjects Who Entered the Treatment Period by Site 7.3.4

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Status of Entrance into the Treatment Period

Stratum:

Site [Site numbers will be used as categories]

Analytical Methods:

(1) Number of Subjects Who Entered the Treatment Period by Site Frequency distributions will be provided for each stratum.

#### 7.3.5 Disposition of Subjects for Follow-up Period

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Study Treatment Administration Status

[Eligible but Not Treated]

Reason for Not Being Treated

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

Completion Status for Follow-up Period

[Completed, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

#### Analytical Methods:

(1) Disposition of Subjects

Frequency distributions will be provided. When calculating percentages for the reasons for not being treated, the total number of subjects not treated will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

(2) Completion Status for Follow-up Period

Frequency distributions will be provided for Completion Status for Follow-up Period(categories of Completed, Ongoing and Prematurely Discontinued).

## 7.3.6 Completion Status for Follow-up Period

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Completion Status for Follow-up Period

[Completed, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

Categories:

Duration of Study after Baseline (days)

Analytical Methods:

(1) Completion Status for Follow-up Period by Duration of Study after Baseline

Frequency distributions will be provided for each category of duration of study after baseline.

# 7.3.7 Disposition of Subjects for Long-Term Follow-up Period

Analysis Set:

All Subjects Who Completed the Follow-up period

## Analysis Variables:

Completion Status for Long-Term Follow-up Period

[Completed/Ongoing, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

#### Analytical Methods:

(1) Disposition of Subjects

Frequency distributions will be provided. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

(2) Completion Status for Long-Term Follow-up Period

Frequency distributions will be provided for Completion Status for Long-Term Follow-up Period (categories of Completed, Ongoing and Prematurely Discontinued).

## 7.3.8 Completion Status for Long-Term Follow-up Period

Analysis Set:

All Subjects Who Completed the Follow-up Period

Analysis Variables:

Completion Status for Long-Term Follow-up Period

[Completed/Ongoing, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

## Categories:

Duration of Study after Baseline (days)

[Min - 547, 548 - 729, 730-911, 912 - Max]

#### **Analytical Methods:**

(1) Completion Status for Long-Term Follow-up Period

Frequency distributions will be provided for each category of duration of study after baseline.

#### **Protocol Deviations and Analysis Sets** 7.3.9

#### 7.3.9.1 Protocol Deviations

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Significant Protocol Deviation

[Entry Criteria, Concomitant Medication, Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria]

Analytical Methods:

(1) Protocol Deviations

Frequency distributions will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

#### 7.3.9.2 Analysis Sets

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Handling of Subjects

[Categories are based on the specifications in Subject Evaluability List]

**Analysis Sets** 

Intention to Treat [Included] Modified Intention to Treat [Included] Per Protocol Set [Included] Safety Analysis Set [Included]

Analytical Methods:

- Subjects Excluded from Analysis Sets

Subjects Excl (2) Analysis Sets Frequer Frequency distributions will be provided. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

## 7.4 Demographic and Other Baseline Characteristics

Analysis Set:

Intention to Treat

Analysis Variables:

Age (years)  $[Min \le - \le 65, 65 \le - \le Max]$ 

Gender [Male, Female]

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$ 

Smoking Classification [Never, Current, Former]

Previous use of Antibiotics [Yes, No]

Previous use of Immunosuppressants [Yes, No]

Previous use of Biologics [Yes, No.

Concomitant Medications [Biologics only, Immunosuppressants only,

Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

Duration of Crohn's Disease (years)

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

[1 IO + 1 EO, 1 IO + 2 EOs, 1 IO + 3 EOs, 2 IOs + 1 EO, 2 IOs + 2 EOs, 2 IOs + 3 EOs]

Topography of Draining EOs at Screening

[0 EO, 1 EO, 2 EOs, 3EOs]

CDAI Total Score at Baseline [Min<= - <150, 150<= - <=220, 220< - <=Max]

Analytical Methods:

(1) Summary of Demographics and Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

## 7.5 Medical History and Concurrent Medical Conditions

Analysis Set:

Safety Analysis Set

Analysis Variables:

Medical History

**Concurrent Medical Conditions** 

Analytical Methods:

- (1) Medical History by System Organ Class and Preferred Term
- (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency. A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

## 7.6 Medication History and Concomitant Medications

Concomitant medications whose start date occurred on or before Week 52 visit, ie, the latest fistula clinical assessment or the latest visit by Day 448, will be summarized.

Analysis Set:

Safety Analysis Set

Analysis Variables:

**Medication History** 

Concomitant Medications

Analytical Methods:

- (1) Medication History by Preferred Medication Name.
- (2) Concomitant Medications That Started and Stopped Prior to Baseline by Preferred Medication Name.
- (3) Concomitant Medications That Started Prior to and Were Ongoing at Baseline by Preferred Medication Name.
- (4) Concomitant Medications That Started After Baseline by Preferred Medication Name.
- (5) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name.

Frequency distributions will be provided. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that preferred medication name.

#### 7.7 **Study Drug Exposure and Compliance**

Analysis Set:

Safety Analysis Set

Analysis Variables:

Total Exposure (mL)

Total Exposure per IOs (mL)

Total Exposure per EOs (mL)

Duration of follow-up after baseline by Week 52 (weeks)

Analytical Methods:

(1) Summary of Total Exposure

Descriptive statistics will be provided.

#### 7.8 **Efficacy Analysis**

#### 7.8.1 **Secondary Endpoints**

Efficacy analysis using data up to Week 52

only and subject to the applicable reins of Use Proportion of Subjects with Combined Remission, Clinical Remission and Response 7.8.1.1 at Week 52

Analysis Set:

Intention to Treat

**Analysis Variables:** 

Combined Remission at Week 52

Clinical Remission at Week 52

Response at Week 52

Analytical Methods:

Frequency distributions will be provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method).

Proportion of Subjects with Relapse at Week 52 in subjects with combined remission at Week 24

Analysis Set:

Intention to Treat

Analysis Variables:

Relapse at Week 52

Analytical Methods:

(1) Number and Percentage of Subjects with Relapse at Week 52
Within the subjects with combined remission at Week 24, frequency distributions will be provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method).

7.8.1.3 Proportion of Subjects with Combined Remission at Week 52 and combined remission at Week 24

Analysis Set:

Intention to Treat

Analysis Variables:

Combined Remission at Week 24 and Week 52

Analytical Methods:

(1) Number and Percentage of Subjects with Combined Remission at Week 24 and Week 52 For the number and percentage of subjects with combined remission at Week 24 and Week 52 as well as the number and percentage of subjects with combined remission at Week 24 and without combined remission at Week 52, frequency distributions will be provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method).

7.8.1.4 Time to Combined Remission, Clinical Remission and Response by Week 52

Analysis Set:

Intention to Treat

Analysis Variables:

Time to Combined Remission by Week 52

Time to Clinical Remission by Week 52

Time to Response by Week 52

Analytical Methods:

For the following time to event analyses, subjects without event will be handled as censor at the date of last fistula clinical assessment.

(1) Summary of Time to Event by Week 52
Frequency distribution of subjects who experienced event and who were censored will be provided. Quartiles of time to event will be estimated using the Kaplan-Meier method.

(2) Kaplan-Meier Plot Kaplan-Meier plot of time to combined remission, clinical remission, and response by

Week 52 will be provided.

#### 7.8.1.5 Time to Relapse by Week 52

Analysis Set:

Intention to Treat

Analysis Variables:

Time to Relapse by Week 52

Analytical Methods:

the applicable terms of Use Within the subjects with combined remission at Week 24, the following analyses will be performed. For the following time to event analyses, subjects without event will be handled as censor at the date of last fistula clinical assessment or last fistula MRI assessment.

- (1) Summary of Time to Event by Week 52 Frequency distribution of subjects who experienced event and who were censored will be provided. Quartiles of time to event will be estimated using the Kaplan-Meier method.
- (2) Kaplan-Meier Plot Kaplan-Meier plot of time to relapse by Week 52 will be provided.

#### PDAI Score 7.8.1.6

Analysis Set:

Intention to Treat

Analysis Variables:

PDAI Total Score

PDAI Domain Scores(Discharge, Pain/restriction of activities, Restriction of Sexual Activity, Type of Perianal Disease, Degree of Induration)

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 40, Week 52

Analytical Methods:

(1) Summary of PDAI Scores and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline for each visit will be provided.

## (2) Mean and Standard Deviation Plots

Mean observed values and changes from baseline will be plotted for each visit with standard deviation bars.

#### 7.8.1.7 *CDAI Score*

Analysis Set:

Intention to Treat

Analysis Variables:

**CDAI Sub Scores** 

Visit:

Baseline, Week 24, Week 52

Analytical Methods:

- (1) Summary of CDAI Scores and Change from Baseline by Visit
  Frequency distribution for categorical variables and descriptive statistics of observed values
  and changes from baseline for each visit will be provided.
- (2) Mean and Standard Deviation Plots

Mean observed values and changes from baseline will be plotted for each visit with standard deviation bars.

#### 7.8.1.8 Van Assche Score

Analysis Set:

Intention to Treat

Analysis Variables:

Van Assche Total Score

Van Assche Domain Scores

Visit:

Baseline, Week 24, Week 52

**Analytical Methods:** 

- (I) Summary of Van Assche Scores and Change from Baseline by Visit Frequency distribution for categorical variables and descriptive statistics of observed values and changes from baseline for each visit for continuous variables will be provided.
- (2) Mean and Standard Deviation Plots
  Mean observed values and changes from baseline will be plotted for each visit with standard deviation bars for continuous variables.

#### 7.8.2 Additional Endpoints

Efficacy analysis using data up to Week 52

7.8.2.1 Timepoint Analysis of Clinical Remission and Response

Analysis Set:

Intention to Treat

Analysis Variables:

Clinical Remission

Response

Visit:

Week 2, Week 4, Week 8, Week 16, Week 24, Week 40, Week 52

Analytical Methods:

The same analysis for the primary endpoint will be performed by visit.

## 7.8.3 Statistical/Analytical Issues

7.8.3.1 Adjustments for Covariates

Not applicable.

# 7.8.3.2 Handling of Dropouts or Missing Data

Values below the lower limit of quantification will be treated as zero when calculating the descriptive statistics. Values above the upper limit of quantification will be treated as the upper limit of quantification when calculating the descriptive statistics.

For combined remission, clinical remission, response

For the primary and secondary analyses of the primary endpoint, the last observation carried forward (LOCF) from the latest earlier post-baseline visit (including an Early Termination Visit prior to Week 24, if applicable) will apply in case of missing clinical assessment at Week 24. In case of missing MRI data at Week 24, LOCF from an Early Termination Visit prior to Week 24 will apply if applicable. In case of no MRI data by Week 24 or no post-baseline clinical assessment, non-response will be imputed. If rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly occur prior to visit 8(Week 24), non-response will be imputed overriding all other imputation conventions.

The handling above for the primary endpoint will also be applied to proportion of subjects with clinical remission at Week 24, proportion of subjects with response at Week 24, proportion of subjects with clinical remission at Week 52, proportion of subjects with clinical remission at Week 52 and proportion of subjects with response at Week 52 (but handling of rescue therapy will not be applied for Week 52).

#### 7.8.3.3 Multicenter Studies

licable Terms of Use Although this study is a multicenter study, treatment-by-center interaction will not be explored since the number of subjects for each center is not sufficient for such exploration.

#### 7.8.3.4 *Multiple Comparison/Multiplicity*

Not applicable.

#### 7.8.3.5 Use of an "Efficacy Subset" of Subjects

In addition to analyses on the primary endpoint using the intention to treat, a secondary analysis will also be performed using the modified intention to treat and the per protocol set to confirm the robustness of the results.

#### Active-Control Studies Intended to Show Equivalence or Non-Inferiority 7.8.3.6 Not applicable.

#### 7.8.3.7 Examination of Subgroups

Efficacy analysis using data up to Week 52

Analysis Set:

Intention to treat

Analysis Variables:

Combined Remission at Week 52

Clinical Remission at Week 52

Response at Week 52

Subgroups:

Age 
$$[Min <= - <= 65, 65 < - <= Max]$$

Male, Female]

Topography of IOs and EOs at Baseline

$$[1 \text{ IO} + 1 \text{ EO}, 1 \text{ IO} + (2 \le \text{EOs}), 2 \text{ IOs} + (1 \le \text{EOs})]$$

Previous use of Antibiotics [Yes, No]

Previous use of Immunosuppressants [Yes, No]

Previous use of Biologics [Yes, No]

ect to the applicable retrins of Use **Concomitant Medications** [Biologics only, Immunosuppressants only, Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

Analytical Methods:

(1) Descriptive Statistics

Frequency distributions will be provided for above each subgroups.

#### 7.9 **Other Outcomes**

Not applicable.

#### 7.10 **Safety Analysis**

Safety analysis using data up to Week 52

#### 7.10.1 **Adverse Events**

TEAEs whose date of onset occurred on or before Week 52 visit, ie, the latest fistula clinical assessment or the latest visit by Day 448, will be summarized.

#### Overview of Treatment-Emergent Adverse Events 7.10.1.1

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

Categories:

Relationship to Study Preatment [Related, Not Related]

Intensity [Mild, Moderate, Severe]

Analytical Methods

The following summaries will be provided.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 2) Relationship of Treatment-Emergent Adverse Events to study treatment (number of events, number and percentage of subjects).
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).

- 4) Treatment-Emergent Adverse Events leading to study discontinuation (number of events, number and percentage of subjects).
- 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
- 6) Relationship of serious Treatment-Emergent Adverse Events to study treatment (number of events, number and percentage of subjects).
- 7) Serious Treatment-Emergent Adverse Events leading to study discontinuation (number of events, number and percentage of subjects).
- 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects).

TEAEs will be counted according to the rules below.

#### Number of subjects

• Summaries for 2) and 6)

A subject with occurrences of TEAE in both categories (ie, Related and Not Related) will be counted once in the Related category.

• Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

• Summaries other than 2), 3), and 6)

A subject with multiple occurrences of TEAE will be counted only once.

#### Number of events

For each summary, the total number of events will be calculated.

## 7.10.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variables:

CEAE

Categories:

Intensity [Mild, Moderate, Severe]

Time of Onset (day) [1 - 57, 58 - 169, 170-281, 282 - Max]

Analytical Methods:

The following summaries will be provided using frequency distribution.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term-
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Study Treatment-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Study Treatment-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over
- (10) Treatment-Emergent Adverse Events of Special Interest by System Organ Class and Preferred Term
- (11) Product Malfunction-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distributions will be provided according to the rules below.

## Number of subjects

• Summary tables other than (5), (6) and (9)

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.

• Summary tables for (5) and (6)

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.

LEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. Percentages will be based on the number of subjects in the safety analysis set

Subgroup Analysis of Treatment-Emergent 1.7

et: a St. sysis se applicable applica

## 7.10.1.3

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

Subgroups:

 $[Min \le - \le 65, 65 \le - \le Max]$ Age

Gender [Male, Female]

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

[1 EO,  $2 \le EOs$ ]

Previous use of Antibiotics

[Yes, No]

Previous use of Immunosuppressants

[Yes, No]

Previous use of Biologics

[Yes, No]

**Concomitant Medications** 

[Biologics only, Immunosuppressants only,

Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

#### Analytical Methods:

The following summaries will be provided for each subgroup using frequency distribution. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT.

1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set for each subgroup.

#### 7.10.1.4 Displays of Pretreatment Events

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

**PTE** 

Analytical Methods:

The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term.
- (2) Serious Pretreatment Events by System Organ Class and Preferred Term.

The frequency distributions will be provided according to the rules below.

## Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

#### 7.10.2 Clinical Laboratory Evaluations

## 7.10.2.1 Hematology and Serum Chemistry

Analysis Set:

Safety Analysis Set

Analysis Variables:

Hematology

Hemoglobin, Hematocrit, Red blood cells count, Mean Corpuscular Volume, Mean Corpuscular Hemoglobin, Mean Corpuscular Hemoglobin Concentration, White blood cells count, differential WBC (Neutrophils, Basophils, Eosinophils, Lymphocytes, Monocytes), Platelet count

Serum Chemistry

C-reactive protein, ALT, AST, Alkaline phosphatase, Gamma-glutamyl transpeptidase, Total bilirubin, Total protein, Glucose, Creatinine, Creatine phosphokinase, Blood urea nitrogen, Potassium, Sodium, Chloride

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 52

## Analytical Methods:

For each variable, summaries (1) to (3) will be provided.

(1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

Be Plots

Plots over time for each subject

The provided of the provide

(2) Case Plots

(3) Summary of Shifts of Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications. cial use only and

#### 7.10.2.2 Urinalysis

## Analysis Set:

Safety Analysis Set

#### Analysis Variables:

Specific Gravity

рН

Glucose

Protein

Occult blood

Ketone body

Bilirubin

Urobilinogen

[+-, +, 2+, 3+]

## Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 52

# Baseline, Week Analytical Methods: For specif

For specific gravity, summaries (1), (2) and (4) will be provided.

For pH, summary (4) will be provided.

For each variable other than specific gravity or pH, summaries (3) and (4) will be provided.

(1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit

3DIE Terms of Use Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Number of Subjects in Categories of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

(4) Summary of Shifts of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

For each urine laboratory test, the laboratory values will be classified as "Low",

"Normal" or "High" for specific gravity and pH, classified as "Normal" or

"Abnormal" for others relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

#### 7.10.3 Vital Signs

Analysis Set:

Safety Analysis Set

Analysis Variables:

Temperature

Systolic Blood Pressure

Diastolic Blood Pressure

Heart Rate

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 40, Week 52

Analytical Methods:

For each variable, summaries (1) and (2) will be provided

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.

#### 7.10.4 Other Observations Related to Safety

7.10.4.1 Donor Specific Antibody

Analysis Set:

Safety Analysis Set

Analysis Variables:

Donor Specific Antibody

[Presence, Absence]
(Categories used in analytical methods (1) and (2))

Presence at baseline and Presence during post-1
Presence at baseline and Absence during besnce at baseline and Presence at baseline and Absence at baseline at ba

Presence at baseline and Absence during post-baseline by Week 52, Absence at baseline and Presence during post-baseline by Week 52, Absence at baseline and Absence during post-baseline by Week 52]

Jaring post-baseline by Week 24

Jaseline after Week 24 by Week 52,

Lesence at baseline and Absence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52,

Presence at baseline and Absence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52,

Presence at baseline and Absence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52,

Absence at baseline and Presence during post-baseline by Week 24 or Presence during post-baseline after Week 24 by Week 52.

Absence at baseline and Presence during post-baseline by Week 24 or Presence during post-baseline after Week 21 by Week 52.

Absence at baseline and Absence during post-baseline after Week 21 by Week 52.

Absence at baseline and Absence during post-baseline after Week 21 by Week 52.

Absence at baseline and Absence during post-baseline after Week 21 by Week 52.

Absence at baseline and Presence during post-baseline after Week 21 by Week 52.

Absence at baseline and Presence during post-baseline by Week 52.

baseline by Week 24]

[Presence during post-baseline by Week 52, Absence during postbaseline by Week 52] (Categories used in analytical method (4))

(Presence/Absence at baseline is results of anti-HLA antibody.)

(Presence/Absence during post-baseline is results of donor specific antibody during postbaseline by Week 24/52, ie, Presence if any positive results during post-baseline by Week 24/52, Absence if no positive results during post-baseline by Week 24/52.)

#### Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 52 Analytical Methods:

(1) Summary of Donor Specific Antibody by Visit Frequency distributions for each visit will be provided

(2) Summary of Shifts of Donor Specific Antibody

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

(3) Number of Subjects in Categories of Donor Specific Antibody

Frequency distributions of results at baseline and during post-baseline by Week 24/52 as well as baseline, during post-baseline by Week 24 and during post-baseline after Week 24 by Week 52 will be provided.

(4) Subgroup Analysis of Efficacy and Safety Endpoints by Donor Specific Antibody

The same analyses of Section 7.8.3.7 and 7.10.1.3 will be conducted for each subgroup of Donor Specific Antibody based on results during post-baseline by Week 52. For the same analyses of Section 7.8.3.7, combined remission at Week 24, clinical remission at Week 24, response at Week 24 will be also analyzed for each subgroup of Donor Specific Antibody based on results during post-baseline by Week 24.

7.10.4.2 Displays of Treatment-Emergent Adverse Events (Japanese)

# Analysis Set:

Safety Analysis Set

Analysis Variables:
TEAF Analytical Methods:

> TEAEs will be summarized in the same way as in section 7.10.1.2 and 7.10.1.3. All summaries will be presented in Japanese.

....y interim analysis. Note, the analysis using data up to Week 24 is the primary analysis for marketing application. Additionally, separate analyses using data up to Week 52 and overall data will be performed after all subjects complete Week 52 and Week 156 respectively.

7.12 Changes in the Statistical Analysis Plan

The analyses in the

specifically and subject to the appropriate appropriat The analyses in the statistical analysis plan do not differ from the analyses specified in the protocol.

Changes from the previous version are listed below.

Page 38, Section 7.10.2.2

**Existing Text** 

Revised Text

Occult blood 
$$[-, +-, +, 2+, 3+]$$
  
Bilirubin  $[-, +-, +, 2+, 3+]$ 

Rationale for Amendment

Modified category of occult blood.

Page 38, Section 7.10.2.2

**Existing Text** 

(4) Summary of Shifts of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

For each urine laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

Revised Text

(4) Summary of Shifts of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

For each urine laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" for specific gravity and pH, classified as "Normal" or

antal of Use applicable Terrison to the applicable of the applicab

# ELECTRONIC SIGNATURES

| | ELECTRONIC SIGNATURES | Zerin Zerin |
|---|---|---|
| Signed by | Meaning of Signature | Server Date |
| Signed by Property of Takeda. For nothing | Biostatistics Approval Biostatistics Approval | (dd-MMM-yyyy HH;main 'UTC') 12-Mar-2021 13:31 UTC |



#### STATISTICAL ANALYSIS PLAN

[Analysis using Data up to Week 156]

the applicable rems of Use STUDY NUMBER: Darvadstrocel-3002

A Phase 3, Multicenter, Open-Label, Uncontrolled Study to Exaliate the Efficacy and Safety of Cx601 in the Treatment of Complex Perianal Fistulas in Adult Patients with Crohn's Disease

Version: 1st
Date: 9 May 2022

Prepared by:

Based on:

Protocol Version: Amendment 5

Protocol Date: 13 April 2021

Properly of Takeda: For non-commercial use only and subject to the applicable Terms of use

## 2.0 TABLE OF CONTENTS

| TABLE OF CONTENTS | 4 | ~ |
|---|---|---|
| 1.0 TITLE PAGE | | 1 |
| 1.1 Approval Signatures | | 2 |
| 2.0 TABLE OF CONTENTS | | 3 |
| List of In-Text Tables | i,C <sup>O</sup> | 5 |
| List of In-Text Figures | | 5 |
| 3.0 LIST OF ABBREVIATIONS | · | 7 |
| 4.0 OBJECTIVES | | 3 |
| 4.1 Primary Objectives | , <sub>1</sub> O | 3 |
| 4.2 Secondary Objectives | | 3 |
| 4.3 Additional Objectives | (0) | 3 |
| 4.4 Study Design | | 3 |
| 5.0 ANALYSIS ENDPOINTS | | 9 |
| 5.1 Primary Endpoint | | 9 |
| 5.2 Secondary Endpoints | | ) |
| 5.3 Safety Endpoints | © | ) |
| 5.4 Additional Endpoints | 1 | 1 |
| | IZE1 | |
| | RESENTATION1 | |
| | 1 | |
| 7.1.1 Study Definitions | 1 | 1 |
| | 12 | |
| 7.1.3 Definition of Study Visit Win | dows1 | 3 |
| 7.1.3.1 Fistula Assessment | 1 | 3 |
| 7.1.3.2 Endpoints Other Than | Fistula Assessment14 | 4 |
| 7.14 Significance Level and Confi | dence Coefficient1 | 7 |
| 7.1.5 Calculation of Combined Rer | nission, Clinical Remission, Response1 | 7 |
| 7.1.6 Calculation of Relapse in Sub | jects with Clinical/Combined Remission18 | 3 |
| 7.2 Analysis Sets | 1 | 9 |
| 7.3 Disposition of Subjects | 20 | ) |
| 7.3.1 Study Information | 20 | ) |
| 7.3.2 Screen Failures | 20 | ) |
| 7.3.3 Subject Eligibility | 2 | 1 |

| 7. | 3.4 Num | ber of Subjects Who Entered the Treatment Period by Site | 21 |
|---|---|---|---|
| 7. | | osition of Subjects for Follow-up Period | |
| 7. | 3.6 Com | pletion Status for Follow-up Period | 22 |
| 7. | 3.7 Disp | osition of Subjects for Long-Term Follow-up Period | .23 |
| 7. | 3.8 Com | pletion Status for Long-Term Follow-up Period ocol Deviations and Analysis Sets Protocol Deviations Analysis Sets aphic and Other Baseline Characteristics History and Concurrent Medical Conditions | 23 |
| 7. | 3.9 Proto | ocol Deviations and Analysis Sets | 24 |
| | 7.3.9.1 | Protocol Deviations | 24 |
| | 7.3.9.2 | Analysis Sets | 24 |
| 7.4 | Demogra | aphic and Other Baseline Characteristics | 25 |
| 7.5 | Medical | History and Concurrent Medical Conditions | 26 |
| 7.6 | | | |
| | Analysis | Set: | 26 |
| 7.7 | Study Di | rug Exposure and Compliance | 27 |
| 7.8 | Efficacy | Analysis | 27 |
| 7. | 8.1 Addi | Set: rug Exposure and Compliance Analysis tional Endpoints Proportion of Subjects with Combined Remission Clinical Remission | 27 |
| | 7.8.1.1 | Proportion of Subjects with Combined Remission, Clinical Remission and Response at Week 104/Week 156 | |
| | 7.8.1.2 | Proportion of Subjects with Relapse at Week 104/Week 156 in subjects with combined remission at Week 52/Week 104 | |
| | 7.8.1.3 | Proportion of Subjects with Combined Remission at Multiple Timepoints | 28 |
| | 7.8.1.4 | Time to Combined Remission, Clinical Remission and Response by Week 104/Week 156. | 29 |
| | 7.8.1.5 | Time to Relapse by Week 104/Week 156 | 29 |
| | 7.8.1.6 | POAI Score | 30 |
| | 7.8.1.7 | CDAI Score | 30 |
| | 7.8.1.8 | Van Assche Score | 31 |
| | 7.8.1.9 | Timepoint Analysis of Clinical Remission and Response | 31 |
| 70 | | stical/Analytical Issues | 31 |
| 1 St | 7.8.2.1 | Adjustments for Covariates | |
| | 7.8.2.2 | Handling of Dropouts or Missing Data | |
| ) ` | 7.8.2.3 | Multicenter Studies | |
| | 7.8.2.4 | Multiple Comparison/Multiplicity | |
| | 7.8.2.5 | Use of an "Efficacy Subset" of Subjects | |
| | 7.8.2.6 | Active-Control Studies Intended to Show Equivalence or Non- | |
| | | Inferiority | 32 |

Propert

| rabie /.a | VISIT WINDOW OF FISTURA MIKE ASSESSMENT | |
|-----------|---------------------------------------------|----|
| Table 7.b | Visit Window of Fistula Clinical Assessment | 14 |
| Table 7.c | Visit Window of PDAI Score | |
| Table 7.d | Visit Window of CDAI Score | 15 |
| Table 7.e | Visit Window of Van Assche Score | 15 |
| Table 7.f | Visit Window of Vital Signs | 16 |
| Table 7.g | Visit Window of Clinical Laboratory Tests | 16 |
| Table 7.h | Visit Window of Anti-donor Antibody Test | 17 |

And set of the state of the sta

#### 3.0 LIST OF ABBREVIATIONS

AE adverse event ALP alkaline phosp

ALP alkaline phosphatase
ALT alanine aminotransferase
AST aspartate aminotransferase
CDAI Crohn's Disease Activity Index
DMEM Dulbecco Modified Eagle's Medium

eASC expanded allogeneic adipose-derived stem cells

ECG electrocardiogram

eCRF electronic case report form
EMA European Medicines Agency

EO External Opening

FDA Food and Drug Administration
GCP Good Clinical Practice

GGT gamma-glutamyl transpeptidase HBsAg hepatitis B virus surface antigen

HBV hepatitis B virus

hCG human chorionic gonadotropin

HCV hepatitis C virus
HSA human serum albumin

ICH International Conference on Harmonisation

IL interleukin

INR international normalized ratio

IO Internal Opening

IRB institutional review board

ITT intention to treat

LOCF last observation carried forward

MedDRA Medical Dictionary for Regulatory Activities
MHLW Ministry of Health, Labour and Welfare

MHRA Medicines and Healthcare products Regulatory Agency

mITT modified intention to treat
MRI magnetic resonance imaging
PCR polymerase chain reaction
PDAI Perianal Disease Activity Index

PMDA Pharmaceuticals and Medical Devices Agency

PPS per protocol set
PTE Pretreatment event
SAE serious adverse event
SAP statistical analysis plan

SUSAR suspected unexpected serious adverse reaction

TEAE treatment-emergent AE
TNF tumor necrosis factor
ULN upper limit of normal
WBC white blood cell

#### 4.0

#### 4.1

To evaluate the efficacy of Cx601 for the treatment of complex perianal fistulas in adult patients with Crohn's disease over 24 weeks.

Secondary Objectives

To evaluate the efficacy of Carte patients with

## 4.2

- patients with Crohn's disease over 52 weeks.
- To evaluate the safety of Cx601 for the treatment of perianal fistulas in adult patients with Crohn's disease over minimum 156 weeks.

#### 4.3 **Additional Objectives**

- To evaluate the absence of clinically relevant alloreactivity.
- To evaluate the effects of Cx601 on Crohn's disease activity and quality of life.

#### 4.4 **Study Design**

This is Phase 3, a multicenter, open-label, uncontrolled study to evaluate the efficacy and safety of Cx601 in the treatment of complex perianal fistulas in adult patients with Crohn's disease.

Subjects with Crohn's disease whose complex perianal fistulas were previously treated and refractory (inadequate response, loss of response or intolerance) to at least one of the following treatments: antibiotics, immunosuppressants or biologics (anti-TNFs, anti-integrin or anti-IL-12/23) will be included in the study. Note that those subjects who are refractory to antibiotics only will be must be less than 25% of all subjects enrolled.

The study will permit continuation of baseline treatments for Crohn's disease in an add-on design (ie, biologics, immunosuppressants, etc.). A total of 20 subjects are planned to be enrolled, and study product, cell suspension containing 120×10<sup>6</sup> cells of eASCs, will be intralesionally injected to all participants. Since this is the first study of Cx601 in Japanese subjects, the enrollment of at least the first 3 subjects will be adjusted not to be administered the study product at the same day.

This study consists of the screening period (approximately 5 weeks prior to study product administration, including the screening visit and the preparation visit), the treatment period (the day of study product administration), the follow-up period (approximately 52 weeks after study product administration), and the long-term follow-up period (from Week 52 to Week 156 or later; for a minimum of 104 weeks). Cx601 will be administrated once on Day 1, and the efficacy and safety of Cx601 will be mainly evaluated in the subsequent 52-week follow-up period. The primary endpoint will be evaluated at Week 24. Additionally, in the long-term

follow-up period after Week 52, a safety follow-up evaluation will be performed for all subjects every 26 weeks (6 months) until Week 156 or later.

In the screening period, a screening visit (Visit 1) to determine a subject's eligibility is scheduled during the period from Day -39 to the day before preparation. All the subjects eligible by the screening will receive fistula curettage and seton placement under anesthesia at the preparation visit (Visit 2: Day -21, done no later than Day -14). Seton(s) placed will be removed on the day of study product administration (Visit 3: Day 1), just before the administration of the study product. Appropriate training for the preparation and the administration will be implemented to standardize the procedures between study sites.

The subjects who meet all the eligibility criteria will visit the study site on Day 1, and receive fistula curettage under anesthesia and an intralesional injection of cell suspension containing  $120\times10^6$  cells of eASCs (Cx601). Thereafter, in follow-up period, the subjects will visit the study site for the clinical assessments including fistula closure at Weeks 2, 4, 8, 16, 24, 40 and 52. Radiological assessments (MRI) of fistula closure will also be performed at Weeks 24 and 52.

Additionally, in the long-term follow-up period, the safety follow-up will be performed on all the subjects (where possible) every 26 weeks (6 months) from a visit in Week 52 through Week 156. This study will be switched to a post-marketing clinical study if Cx601 is approved before the study completion.

A schematic study design is shown in Figure 4.a.

SCREENING FOLLOW-UP Fistula clinical [Preparation Visit] **Gurettage &** assessment Curettage with study Product seton placement [Screening Visit] VISIT 1 VISIT 3 VISIT 4 VISIT 5 VISIT 6 VISIT 7 VISIT 8 VISIT 9 VISIT 10 W16 W24 W40 W52 Primary Endpoint Fistula clinical 8 MRI assessmen MRI assessment LONG-TERM FOLLOW-UP continued from W52 VISIT 10 VISIT 11 VISIT 12 VISIT 13 VISIT 14 W130 W156

Figure 4.a Schematic Study Design

#### 5.0 ANALYSIS ENDPOINTS

## 5.1 Primary Endpoint

Proportion of subjects with combined remission at Week 24.

## 5.2 Secondary Endpoints

#### Efficacy analysis using data up to Week 24:

- Proportion of subjects with clinical remission at Week 24.
- Proportion of subjects with response at Week 24.
- Time to clinical remission by Week 24.
- Time to response by Week 24.
- Proportion of subjects with relapse at Week 24 in subjects with clinical remission at previous visit.
- Time to relapse by Week 24 in subjects with clinical remission at previous visit.
- PDAI score (including total score, discharge sub-score and pain sub-score) up to Week 24.
- CDAI score up to Week 24.
- Van Assche score up to Week 24.

## Efficacy analysis using data up to Week 52:

- Proportion of subjects with combined remission at Week 52.
- Proportion of subjects with clinical remission at Week 52.
- Proportion of subjects with response at Week 52.
- Time to combined remission by Week 52.
- Time to clinical remission by Week 52.
- Time to response by Week 52.
- Proportion of subjects with relapse at Week 52 in subjects with combined remission at Week 24.
- Time to relapse by Week 52 in subjects with combined remission at Week 24.
- PDAI score (including total score, discharge sub-score and pain sub-score) up to Week 52.
- CDAI score up to Week 52.
- Van Assche score up to Week 52.

## 5.3 Safety Endpoints

- Adverse events (AEs) including serious adverse events (SAEs) and AEs of special interest.
- Product malfunctions.
- Physical examination findings.
- Vital signs (heart rate, blood pressure, body temperature).
- Clinical laboratory test results (serum chemistry, hematology and urinalysis).

### 5.4 Additional Endpoints

• Presence/absence of anti-donor antibody.

### 6.0 DETERMINATION OF SAMPLE SIZE

The planned sample size is 20 based on feasibility. However, this study has at least 94% probability to show a proportion of subjects with combined remission of 35% or more given an expected proportion of subjects with combined remission of 50% based on Week 24 results in the Cx601-0302 study.

# 7.0 METHODS OF ANALYSIS AND PRESENTATION

### 7.1 General Principles

### 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE) An adverse event whose date of onset occurs on or after receiving study treatment.
- Pretreatment event (PTE): Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to study treatment administration.
- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles.
- Duration of study after baseline (days): Date of last visit/contact date of study treatment administration + 1.
  - If subject is ongoing, date of last visit/contact will be imputed by date of data cut off.
- Duration of follow-up after baseline by Week 156 (weeks): (Date of the latest fistula clinical assessment or the latest visit date of study treatment administration + 1)/7.
- Duration of Crohn's Disease (years): (Date of informed consent date of Crohn's disease diagnosis)/365.25.
  - (If month of diagnosis is missing, month will be replaced with January. If day of diagnosis is missing, day will be replaced with 1<sup>st</sup>.)
- Combined remission: Defined as the clinically confirmed closure of all treated external openings that were draining at the screening despite gentle finger compression, and absence of collections >2 cm in the treated fistulas which is confirmed by the central MRI assessment

(a collection >2 cm is considered as present if at least two out of the 3 dimensions centrally assessed are >2 cm in any of fistula tract).

- Clinical remission: Defined as the clinically confirmed closure of all treated external openings that were draining at the screening despite gentle finger compression.
- Response: Defined as the clinically confirmed closure of at least 50% of all treated external openings that were draining at the screening despite gentle finger compression. Note: Clinically confirmed closure of at least 50% is defined as 1 closure for subjects with 1 baseline external opening, 1 or 2 closures for subjects with 2 baseline external openings, and 2 or 3 closures for subjects with 3 baseline external openings.
- Relapse: Defined as the clinically confirmed reopening of any of the treated external openings with active drainage, or the development of a collection >2 cm in the treated fistulas confirmed by central MRI assessment (a collection >2 cm is considered as present if at least two out of the 3 dimensions centrally assessed are >2 cm in any of fistula tract).
- Time to combined remission/clinical remission/response (days): The time from the study treatment administration to the first visit by which combined remission/clinical remission/response is observed.
   For combined remission, date is the latest of fistula MRI assessment and fistula clinical assessment.
- Time to relapse (days): The time from the first visit which clinical remission is observed to the first visit by which relapse is observed.
   (Time to relapse by Week 104/Week 156 in subjects who achieved combined remission at Week 52/Week 104 is defined as "the time from the combined remission at Week 52/Week 104 to the first visit by which relapse is observed.)
- Presence/Absence of donor specific antibody: Results for each post-baseline visit will be
  presence when at least one of donor specific antibody tests (Class I and/or Class II) is
  presence, otherwise results will be absence. A result at baseline will represent
  presence/absence of anti-HLA Class I and Class II antibody.
- CDAI total score: CDAI total score and body weight will be cut-off by -10, i.e. score below 10 will be treated as -10.

### 7.1,2 Definition of Study Days

The following definitions and calculation formulas will be used.

• Study Day: The day before study treatment administration will be defined as Study Day -1 and the day of the study treatment administration will be defined as Study Day 1. If the date of the observation is on the same date or after the day of the study treatment administration, Study Day will be calculated relative to Study Day 1. Otherwise, Study Day will be calculated relative to Study Day -1.

### 7.1.3 Definition of Study Visit Windows

When calculating Study Day relative to a reference date (ie, study treatment administration [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

### 7.1.3.1 Fistula Assessment

All evaluable data (ie, non-missing data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the largest Study Day will be used.

Table 7.a Visit Window of Fistula MRI Assessment

| Week 24 Week 52 Week 104 Week 156 Week 24(LOCF) Week 52(LOCF) | Study Day: Study Day: Study Day: Study Day: Study Day: Study Day: Study Day: | | Time Interval (days) Study Day - Day Before Preparation 2 - 198 199 - 448 |
|---|---|---|---|
| Week 24 Week 52 Week 104 Week 156 Week 24(LOCF) | Study Day: Study Day: Study Day: Study Day: | Day Before<br>Preparation<br>169<br>365 | - Day Before Preparation<br>2 - 198 |
| Week 24 Week 52 Week 104 Week 156 Week 24(LOCF) | Study Day:<br>Study Day:<br>Study Day: | Preparation<br>169<br>365 | 2 - 198 |
| Week 52 Week 104 Week 156 Week 24(LOCF) | Study Day:<br>Study Day: | 365 | |
| Week 104 Week 156 Week 24(LOCF) | Study Day: | ~ _ | 199 - 448 |
| Week 156<br>Week 24(LOCF) | | 729 | |
| Week 24(LOCF) | Study Day: | 5 129 | 449 - 812 |
| | Stady Buy | 1093 | 813 - |
| Week 52(LOCE) | Study Day: | | 2 - 198 |
| week 32(LOCF) | Study Day: | | 2 - 448 |
| Week 104(LOCF) | Study Day: | | 2 - 812 |
| Week 156(LOCF) | Study Day: | | 2 - |
| Week 104(LOCF) Week 156(LOCF) | | | |

Table 7.b Visit Window of Fistula Clinical Assessment

| | Scheduled Study Day | | Time Interval (days) |
|---|---|---|---|
| Visit | (da | ys) | Study Day |
| Baseline | Study Day: | Day Before<br>Preparation | - Day Before Preparation |
| Week 2 | Study Day: | 15 | 2 - 22 |
| Week 4 | Study Day: | 29 | 23 - 43 |
| Week 8 | Study Day: | 57 | 44 - 85 |
| Week 16 | Study Day: | 113 | 86 - [41 |
| Week 24 | Study Day: | 169 | 142 - 198 |
| Week 40 | Study Day: | 281 | 199 - 323 |
| Week 52 | Study Day: | 365 | 324 - 448 |
| Week 104 | Study Day: | 729 | 449 - 812 |
| Week 156 | Study Day: | 1093 | 813 - |
| Week 2(LOCF) | Study Day: | 39 | 2 - 22 |
| Week 4(LOCF) | Study Day: | 200 | 2 - 43 |
| Week 8(LOCF) | Study Day: | 12,0 | 2 - 85 |
| Week 16(LOCF) | Study Day: | 20/3 | 2 - 141 |
| Week 24(LOCF) | Study Day: | 0, | 2 - 198 |
| Week 40(LOCF) | Study Day: | (5) | 2 - 323 |
| Week 52(LOCF) | Study Day: | <u> </u> | 2 - 448 |
| Week 104(LOCF) | Study Day: | | 2 - 812 |
| Week 156(LOCF) | Study Day: | | 2 - |

# 7.1.3.2 Endpoints Other Than Fistula Assessment

All evaluable data (ie non-missing data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day for others, the later observation will be used.

Table 7.c Visit Window of PDAI Score

| Darvadstrocel-3002<br>Statistical Analysis Plan | | | | <br>9 May 2022 |
|---|---|---|---|---|
| Γable 7.c Visit W | Vindow of PDAI Sco | re | | O. T. |
| Visit | Scheduled Study | Day _ | Time Interval<br>(days) | 9 May 2022 9 May 2022 On Phicable |
| Baseline | (days) Study Day: | 1 | -39 - 1 | |
| Week 2 | Study Day: | 15 | 2 - 22 | - |
| Week 4 | Study Day: | 29 | 23 - 43 | - |
| Week 8 | Study Day: | 57 | 44 - 85 | - 2011 |
| Week 16 | Study Day: | 113 | 86 - 141 | |
| Week 24 | Study Day: | 169 | 142 - 198 | - CO |
| Week 40 | Study Day: | 281 | 199 - 323 | <b>₹</b> 7 |
| Week 52 | Study Day: | 365 | 324 - 448 | - |
| Week 104 | Study Day: | 729 | 449 - 812 | - |
| Week 156 | Study Day: | 1093 | 813 - | - |

**Visit Window of CDAI Score** Table 7.d

| | Scheduled Study I | Day _ | Time Interval<br>(days) |
|----------|-------------------|-------|-------------------------|
| Visit | (days) | | Study Day |
| Baseline | Study Day: | 1 | -39 - 1 |
| Week 24 | Study Day: | 169 | 2 - 198 |
| Week 52 | Study Day: | 365 | 199 - 448 |
| Week 156 | Study Day: | 1093 | 449 - |

Visit Window of Van Assche Score Table 7.e

| K01 | Scheduled Study | Day | Time Interval<br>(days) |
|----------|-----------------|------|-------------------------|
| Visit | (days) | | Study Day |
| Baseline | Study Day: | -35 | -391 |
| Week 24 | Study Day: | 169 | 1 - 198 |
| Week 52 | Study Day: | 365 | 199 - 448 |
| Week 156 | Study Day: | 1093 | 449 - |

Visit Window of Vital Signs Table 7.f

| Darvadstrocel-3002<br>Statistical Analysis Plan | | | | 9 May 2022 |
|---|---|---|---|---|
| Table 7.f Visit V | Vindow of Vital Signs | 1 | | |
| <b>V</b> /::4 | Scheduled Study | Day . | Time Interval<br>(days) | SINS |
| Visit<br>Baseline | (days) Study Day: | 1 | -39 - 1 | |
| Week 2 | Study Day: | 15 | 2 - 22 | - |
| Week 4 | Study Day: | 29 | 23 - 43 | - |
| Week 8 | Study Day: | 57 | 44 - 85 | - |
| Week 16 | Study Day: | 113 | 86 - 141 | - 08, |
| Week 24 | Study Day: | 169 | 142 - 198 | - C |
| Week 40 | Study Day: | 281 | 199 - 323 | <i>₹</i> 3 |
| Week 52 | Study Day: | 365 | 324 - 448 | _ |
| Week 78 | Study Day: | 547 | 449 - 638 | _ |
| Week 104 | Study Day: | 729 | 639 812 | = |
| Week 130 | Study Day: | 911 | 813 - 1002 | - |
| Week 156 | Study Day: | 1093 | 1003 - | - |

Visit Window of Clinical Laboratory Tests Table 7.g

| | Scheduled Study | Day _ | Time Interval<br>(days) |
|----------|-----------------|-------|-------------------------|
| Visit | (days) | | Study Day |
| Baseline | Study Day: | 1 | -39 - 1 |
| Week 2 | Study Day: | 15 | 2 - 22 |
| Week 4 | Study Day: | 29 | 23 - 43 |
| Week 8 | Study Day: | 57 | 44 - 85 |
| Week 16 | Study Day: | 113 | 86 - 141 |
| Week 24 | Study Day: | 169 | 142 - 198 |
| Week 52 | Study Day: | 365 | 199 - 448 |
| Week 104 | Study Day: | 729 | 449 - 812 |
| Week 156 | Study Day: | 1093 | 813 - |

Week 156

| Darvadstrocel-3002<br>Statistical Analysis Plan | | | | <br>9 May 2022 |
|---|---|---|---|---|
| Table 7.h Visit W | indow of Anti-dono | r Antibody | y Test | |
| | Scheduled Study | Day | Time Interval<br>(days) | e applicable retrins of |
| Visit | (days) | | Study Day | <b>√</b> ⊗′ |
| Baseline | Study Day: | 1 | -39 - 1 | |
| Week 2 | Study Day: | 15 | 2 - 22 | |
| Week 4 | Study Day: | 29 | 23 - 43 | - 'iC' |
| Week 8 | Study Day: | 57 | 44 - 85 | - 0'S'. |
| Week 16 | Study Day: | 113 | 86 - 141 | |
| Week 24 | Study Day: | 169 | 142 - 198 | <u> </u> |
| Week 52 | Study Day: | 365 | 199 - 448 | |
| Week 104 | Study Day: | 729 | 449 - 812 | - |

Table 7.h Visit Window of Anti-donor Antibody Test

### Significance Level and Confidence Coefficient

Confidence coefficient: 90% (two-sided), 95% (two-sided).

Study Day:

### 7.1.5 Calculation of Combined Remission, Clinical Remission, Response

Combined Remission at Week 24(Primary endpoint)

Fistula MRI assessment at Week 24(LOCF) and fistula clinical assessment at Week 24(LOCF) will be used when combined remission at Week 24 is calculated based on the definition of section 7.1.1.

1093

If either of the two is missing, non-remission will be imputed.

If a subject received rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly prior to visit 8(Week 24) will be handled as non-remission.

- Clinical Remission, Response at Week 24(Secondary endpoint). Fistula clinical assessment at Week 24(LOCF) will be used when clinical remission or response at Week 24 is calculated based on the definition of section 7.1.1. If fistula clinical assessment is missing, non-remission(non-response) will be imputed. If a subject received rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly prior to visit 8(Week 24) will be handled as non-remission.
- Combined Remission at Week 52(Secondary endpoint). Fistula MRI assessment at Week 52(LOCF) and fistula clinical assessment at Week 52(LOCF) will be used when combined remission at Week 52 is calculated based on the definition of section 7.1.1.

If either of the two is missing, non-remission will be imputed.

- Clinical Remission, Response at Week 52(Secondary endpoint).
   Fistula clinical assessment at Week 52(LOCF) will be used when clinical remission or response at Week 52 is calculated based on the definition of section 7.1.1.
   If fistula clinical assessment is missing, non-remission(non-response) will be imputed.
- Combined Remission at Week 104/Week 156(Additional endpoint).
   Fistula MRI assessment at Week 104(LOCF)/Week 156(LOCF) and fistula clinical assessment at Week 104(LOCF)/156(LOCF) will be used when combined remission at Week 104/Week 156 are calculated based on the definition of section 7.1.1.
   If either of the two is missing, non-remission will be imputed.
- Clinical Remission, Response at Week 104/Week 156(Additional endpoint).
   Fistula clinical assessment at Week 104(LOCF)/Week 156(LOCF) will be used when clinical remission or response at Week 104/Week 156 are calculated based on the definition of section 7.1.1.

   If fistula clinical assessment is missing, non-remission(non-response) will be imputed.
- Clinical Remission, Response for Time Point Analysis(Additional endpoint).
   Fistula clinical assessment at each analysis visit after baseline in Table 7.b other than LOCF will be used when clinical remission or response for each time point analysis is calculated based on the definition of section 7.1.1.
   If fistula clinical assessment is missing, it will be handled as missing.

### 7.1.6 Calculation of Relapse in Subjects with Clinical/Combined Remission

• Relapse at Week 24 in subjects with clinical remission at previous visit.

The first clinical remission date before Day 198 will be identified. Per subject with clinical remission above, subject will be defined as relapsed if there is a fistula MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the first clinical remission and by Day 198 based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

• Relapse at Week 52 in subjects with combined remission at Week 24.

The combined remission date at Week 24(latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 198, the subject will be defined as relapsed if there is a MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the combined remission date and by Day 448 based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

• Relapse at Week 104 in subjects with combined remission at Week 52.

The combined remission date at Week 52(latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 448, the subject will be defined as relapsed if there is a MRI assessment of >2 cm or a clinical assessment of reopening of external openings

Day 812 based on the definition of will be identified. Per subject with combined remission above and who have at least one fietal melapsed if there is a MRI assessment of >2 cm or openings with active drains. section 7.1.1. Otherwise the subject will be defined as non-relapsed.

Relapse at Week 156 in subjects with combined remission at Week 24.

The combined remission date at Week 24 (latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 198, the subject will be defined as relapsed if there is a MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the combined remission date based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

Relapse at Week 156 in subjects with combined remission at Week 52.

The combined remission date at Week 52 (latest date of MRI and clinical assessment, LOCF) will be identified. Per subject with combined remission above and who have at least one fistula MRI assessment or fistula clinical assessment after Day 448, the subject will be defined as relapsed if there is a MRI assessment of >2 cm or a clinical assessment of reopening of external openings with active drainage after the combined remission date based on the definition of section 7.1.1. Otherwise the subject will be defined as non-relapsed.

### 7.2 **Analysis Sets**

- Intention to treat (ITT): All subjects who have enrolled into treatment period.
- Modified intention to treat (mITT): All subjects who have received the study treatment and whose primary efficacy endpoint is evaluable.
- Per protocol set (PPS): All subjects who have completed the minimum protocol-specified procedures without any major protocol deviations (ie, subjects who met the following criteria will be excluded from the PPS).
  - Subjects who did not meet inclusion criteria #3, #5, #6, or #7.
  - Subjects who met exclusion criteria #1, #2, #3, #4, #5, #6, #7, #8, #9, #10, #11, #21, #23, #24, #25, or #27.

- Subjects who have violated the rules for medications and treatments specified in section 7.3 of the protocol prior to visit 8(Week 24).
- Subjects who have violated the rules for rescue therapy specified in section 7.4 of the protocol prior to visit 8(Week 24).
- Subjects who received less than 24 mL of the study treatment.
- Subjects who did not have either fistula MRI assessment or fistula clinical assessment 45 days prior to or post Study Day 169.
- Safety analysis set:

All subjects who have received the study treatment.

### 7.3 Disposition of Subjects

### 7.3.1 Study Information

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version

WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical Methods:

(1) Study Information

Study information shown in the analysis variables section will be provided.

### 7.3.2 Screen Failures

Analysis Set:

All Subjects Who Did Not Enter the Treatment Period

Analysis Variables:

Age (years)

Gender [Male, Female]

### Analytical Methods:

(1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

### 7.3.3 Subject Eligibility

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

Eligibility Status

[Eligible for Entrance into the Treatment Period, Not Eligible for Entrance into the Treatment Period]

Primary Reason for Subject Not Being Eligible

[Death, Adverse Event, Screen Failure, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

### Analytical Methods:

(1) Eligibility for Entrance into the Treatment Period

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will be used as the denominator.

### 7.3.4 Number of Subjects Who Entered the Treatment Period by Site

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Status of Entrance into the Treatment Period [Entered]

Stratum:

Site [Site numbers will be used as categories]

Analytical Methods:

(1) Number of Subjects Who Entered the Treatment Period by Site

Frequency distributions will be provided for each stratum.

### 7.3.5 Disposition of Subjects for Follow-up Period

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Study Treatment Administration Status

[Eligible but Not Treated]

Reason for Not Being Treated

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

Completion Status for Follow-up Period

[Completed, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

Analytical Methods:

(1) Disposition of Subjects

Frequency distributions will be provided. When calculating percentages for the reasons for not being treated, the total number of subjects not treated will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

(2) Completion Status for Follow-up Period

Frequency distributions will be provided for Completion Status for Follow-up Period (categories of Completed, Ongoing and Prematurely Discontinued).

### 7.3.6 Completion Status for Follow-up Period

Analysis Set.

All Subjects Who Entered the Treatment Period

Analysis Variables:

Completion Status for Follow-up Period

[Completed, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

### Categories:

Duration of Study after Baseline (days)

[Min - 57, 58 - 169, 170-281, 282 - Max]

### **Analytical Methods:**

Je Terms of Use (1) Completion Status for Follow-up Period by Duration of Study after Baseline Frequency distributions will be provided for each category of duration of study after baseline. Joject to the apr

### 7.3.7 Disposition of Subjects for Long-Term Follow-up Period

Analysis Set:

All Subjects Who Completed the Follow-up period

Analysis Variables:

Completion Status for Long-Term Follow-up Period

[Completed, Prematurely Discontinued]

Reason for Discontinuation

[Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Otherl

### **Analytical Methods:**

(1) Disposition of Subjects

Frequency distributions will be provided. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

(2) Completion Status for Long-Term Follow-up Period

Frequency distributions will be provided for Completion Status for Long-Term Follow-up Period (categories of Completed and Prematurely Discontinued).

# 7.3.8 Completion Status for Long-Term Follow-up Period

Analysis Set:

All Subjects Who Completed the Follow-up Period

Analysis Variables:

Completion Status for Long-Term Follow-up Period

[Completed, Prematurely Discontinued]

Reason for Discontinuation

applicable Terms of Use [Death, Adverse Event, Lack of Efficacy, Protocol Deviation, Lost to Follow-up, Withdrawal by Subject, Study Terminated by Sponsor, Pregnancy, Other]

### Categories:

Duration of Study after Baseline (days)

[Min - 547, 548 - 729, 730-911, 912 - Max]

### Analytical Methods:

(1) Completion Status for Long-Term Follow-up Period

Frequency distributions will be provided for each category of duration of study after baseline.

### 7.3.9 Protocol Deviations and Analysis Sets

### 7.3.9.1 Protocol Deviations

Analysis Set:

Analysis Variables:

All Subjects Who Entered the Treatment Period of Significant Protocol Deviation [Entry Criteria, Concomitant Medication, Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria]

### Analytical Methods:

(1) Protocol Deviations

Frequency distributions will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

### 7.3.9.2 Analysis Sets

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variables:

Handling of Subjects

[Categories are based on the specifications in Subject Evaluability List]

### **Analysis Sets**

Intention to Treat [Included] Modified Intention to Treat [Included] Per Protocol Set [Included] Safety Analysis Set [Included]

### Analytical Methods:

- (1) Subjects Excluded from Analysis Sets
- (2) Analysis Sets

Re applicable reims of Use ver-Frequency distributions will be provided. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

### Demographic and Other Baseline Characteristics 7.4

Analysis Set:

Intention to Treat

Analysis Variables:

Age (years)

[Male, Female] Gender

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$ 

Smoking Classification [Never, Current, Former]

Previous use of Antibiotics [Yes, No]

Previous use of Immunosuppressants [Yes, No]

Previous use of Biologics [Yes, No]

Concomitant Medications [Biologics only, Immunosuppressants only,

Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

Duration of Crohn's Disease (years)

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

[1 IO + 1 EO, 1 IO + 2 EOs, 1 IO + 3 EOs, 2 IOs + 1 EO, 2 IOs + 2 EOs, 2 IOs + 3 EOs]

Topography of Draining EOs at Screening

[0 EO, 1 EO, 2 EOs, 3EOs]

CDAI Total Score at Baseline

Analytical Methods:

(1) Summary of Demographics and Baseline Characteristics

or controlling and subject to the app Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

### 7.5 **Medical History and Concurrent Medical Conditions**

Analysis Set:

Safety Analysis Set

**Analysis Variables:** 

Medical History

**Concurrent Medical Conditions** 

Analytical Methods:

- (1) Medical History by System Organ Class and Preferred Term
- (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency. A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

### 7.6 **Medication History and Concomitant Medications**

Analysis Set:

Safety Analysis Set

Analysis Variables:

**Medication History** 

**Concomitant Medications** 

Analytical Methods:

(1) Medication History by Preferred Medication Name

- (2) Concomitant Medications That Started and Stopped Prior to Baseline by Preferred Medication Name
- (3) Concomitant Medications That Started Prior to and Were Ongoing at Baseline by Preferred Medication Name
- (4) Concomitant Medications That Started After Baseline by Preferred Medication Name
- (5) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name

Frequency distributions will be provided. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that Jise Orlly and subject preferred medication name.

### 7.7 **Study Drug Exposure and Compliance**

Analysis Set:

Safety Analysis Set

Analysis Variables:

Total Exposure (mL)

Total Exposure per IOs (mL)

Total Exposure per EOs (mL)

Duration of follow-up after baseline by Week 156 (weeks)

Analytical Methods:

(1) Summary of Total Exposure

Descriptive statistics will be provided.

### **Efficacy Analysis** 7.8

### **Additional Endpoints**

Efficacy analysis using data up to Week 156

7.8.1.1 Proportion of Subjects with Combined Remission, Clinical Remission and Response at Week 104/Week 156

Analysis Set:

Intention to Treat

### Analysis Variables:

Combined Remission at Week 104/Week 156

Clinical Remission at Week 104/Week 156

Response at Week 104/Week 156

### Analytical Methods:

Frequency distributions will be provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method).

7.8.1.2 Proportion of Subjects with Relapse at Week 104/Week 156 in subjects with combined remission at Week 52/Week 104

### Analysis Set:

Intention to Treat

Analysis Variables:

Relapse at Week 104/Week 156

Analytical Methods:

- (1) Number and Percentage of Subjects with Relapse at Week 104/Week 156 Within the subjects with combined remission at Week 52/Week 104, frequency distributions will be provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method).
- 7.8.1.3 Proportion of Subjects with Combined Remission at Multiple Timepoints

### Analysis Set:

Intention to Treat

Analysis Variables:

Combined Remission at Week 24, Week 52 and Week 104

Combined Remission at Week 24, Week 52, Week 104 and Week 156

Combined Remission at Week 52 and Week 104

Combined Remission at Week 52, Week 104 and Week 156

### Analytical Methods:

Number and Percentage of Subjects with Combined Remission at Multiple Timepoints For the number and percentage of subjects with combined remission at multiple timepoints, frequency distributions will be provided with proportion and the two-sided 90% and 95% confidence intervals(Wald's method). Denominator of the percentage will be the number of subjects who have assessment in Week 104 or Week 156 time window range(i.e. Day 449 or Day 813 -).

# applicable Terms of Use 7.8.1.4 Time to Combined Remission, Clinical Remission and Response by Week 104/Week 156

### Analysis Set:

Intention to Treat

### Analysis Variables:

Time to Combined Remission by Week 104/Week 156

Time to Clinical Remission by Week 104/Week 156

Time to Response by Week 104/Week 156

### Analytical Methods:

For the following time to event analyses, subjects without event will be handled as censor at the date of last fistula clinical assessment.

- (1) Summary of Time to Event by Week 104/Week 156 Frequency distribution of subjects who experienced event and who were censored will be provided. Quartiles of time to event will be estimated using the Kaplan-Meier method.
- (2) Kaplan-Meier Plot Kaplan-Meier plot of time to combined remission, clinical remission, and response by Week 104/Week 156 will be provided.

### 7.8.1.5 Time to Relapse by Week 104/Week 156

### Analysis Set:

Intention to Treat

### Analysis Variables:

Time to Relapse by Week 104/Week 156

### Analytical Methods:

Within the subjects with combined remission at Week 52/Week 104, the following analyses will be performed. For the following time to event analyses, subjects without event will be handled as censor at the date of last fistula clinical assessment or last fistula MRI assessment.

- (1) Summary of Time to Event by Week 104/Week 156 Frequency distribution of subjects who experienced event and who were censored will be provided. Quartiles of time to event will be estimated using the Kaplan-Meier method.
- (2) Kaplan-Meier Plot Kaplan-Meier plot of time to relapse by Week 104/Week 156 will be provided.

### 7.8.1.6 *PDAI Score*

Analysis Set:

Intention to Treat

Analysis Variables:

**PDAI Total Score** 

PDAI Domain Scores(Discharge, Pain/restriction of activities, Restriction of Sexual Activity, Type of Perianal Disease, Degree of Induration)

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 40, Week 52, Week 104, Week 156

Analytical Methods:

- (1) Summary of PDAI Scores and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline for each visit will be provided.
- (2) Mean and Standard Deviation Plots
  Mean observed values and changes from baseline will be plotted for each visit with standard deviation bars.

### 7.8.1.7 *CDAI Score*

Analysis Set:

Intention to Treat

Analysis Variables:

CDAI Sub Scores

Visit:

Baseline, Week 24, Week 52, Week 156

Analytical Methods:

- (1) Summary of CDAI Scores and Change from Baseline by Visit
  Frequency distribution for categorical variables and descriptive statistics of observed values and changes from baseline for each visit will be provided.
- (2) Mean and Standard Deviation Plots

  Mean observed values and changes from baseline will be plotted for each visit with standard deviation bars.

### 7.8.1.8 Van Assche Score

Analysis Set:

Intention to Treat

Analysis Variables:

Van Assche Total Score

Van Assche Domain Scores

Visit:

Baseline, Week 24, Week 52, Week 156

Analytical Methods:

- to the applicable terms of Use applicable terms of Use (1) Summary of Van Assche Scores and Change from Baseline by Visit Frequency distribution for categorical variables and descriptive statistics of observed values and changes from baseline for each visit for continuous variables will be provided.
- (2) Mean and Standard Deviation Plots Mean observed values and changes from baseline will be plotted for each visit with standard deviation bars for continuous variables.

### 7.8.1.9 Timepoint Analysis of Clinical Remission and Response

Analysis Set:

Intention to Treat

Analysis Variables:

Clinical Remission

Response

Visit:

Week 2, Week 4, Week 8, Week 16, Week 24, Week 40, Week 52, Week 104, Week 156 Analytical Methods:

The same analysis for the primary endpoint will be performed by visit.

# Statistical/Analytical Issues

7.8.2.1 Adjustments for Covariates

Not applicable.

### 7.8.2.2 Handling of Dropouts or Missing Data

Values below the lower limit of quantification will be treated as zero when calculating the descriptive statistics. Values above the upper limit of quantification will be treated as the upper limit of quantification when calculating the descriptive statistics.

For combined remission, clinical remission, response

For the primary and secondary analyses of the primary endpoint, the last observation earried forward (LOCF) from the latest earlier post-baseline visit (including an Early Termination Visit prior to Week 24, if applicable) will apply in case of missing clinical assessment at Week 24. In case of missing MRI data at Week 24, LOCF from an Early Termination Visit prior to Week 24 will apply if applicable. In case of no MRI data by Week 24 or no post-baseline clinical assessment, non-response will be imputed. If rescue therapy which is not allowed in section 7.4 of the protocol or medications which could affect fistula closure directly occur prior to visit 8(Week 24), non-response will be imputed overriding all other imputation conventions.

The handling above for the primary endpoint will also be applied to proportion of subjects with clinical remission at Week 24, proportion of subjects with response at Week 24, proportion of subjects with clinical remission at Week 52, proportion of subjects with clinical remission at Week 52, proportion of subjects with combined remission at Week 104, proportion of subjects with clinical remission at Week 104, proportion of subjects with combined remission at Week 156, proportion of subjects with clinical remission at Week 156 and proportion of subjects with response at Week 156 (but handling of rescue therapy will not be applied for Week 52, Week 104, or Week 156).

### 7.8.2.3 Multicenter Studies

Although this study is a multicenter study, treatment-by-center interaction will not be explored since the number of subjects for each center is not sufficient for such exploration.

### 7.8.2.4 Multiple Comparison/Multiplicity

Not applicable,

## 7.8.2.5 Use of an "Efficacy Subset" of Subjects

In addition to analyses on the primary endpoint using the intention to treat, a secondary analysis will also be performed using the modified intention to treat and the per protocol set to confirm the robustness of the results.

7.8.2.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

Not applicable.

### 7.8.2.7 Examination of Subgroups

Efficacy analysis using data up to Week 104/Week 156

Analysis Set:

Intention to treat

Analysis Variables:

Combined Remission at Week 104/Week 156

Clinical Remission at Week 104/Week 156

Response at Week 104/Week 156

Subgroups:

Age 
$$[Min \le - \le 65, 65 \le - \le Max]$$

Gender [Male, Female]

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

$$[1 \text{ IO} + 1 \text{ EO}, 1 \text{ IO} + (2 \le \text{EOs}), 2 \text{ IOs} + (1 \le \text{EOs})]$$

Previous use of Antibiotics

[Yes, No]

Previous use of Immunosuppressants [Yes, No]

Previous use of Biologics

[Yes, No]

Concomitant Medications [Biologics only, Immunosuppressants only, Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

Analytical Methods:

(1) Descriptive Statistics

Frequency distributions will be provided for above each subgroups.

### 7.9 Other Outcomes

Not applicable.

### 7.10 Safety Analysis

Safety analysis using data up to Week 156

### 7.10.1 Adverse Events

7.10.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

Categories:

Relationship to Study Treatment [Related, Not Related]

Intensity [Mild, Moderate, Severe]

Analytical Methods:

The following summaries will be provided.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 2) Relationship of Treatment-Emergent Adverse Events to study treatment (number of events, number and percentage of subjects).
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 4) Treatment-Emergent Adverse Events leading to study discontinuation (number of events, number and percentage of subjects).
  - 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 6) Relationship of serious Treatment-Emergent Adverse Events to study treatment (number of events, number and percentage of subjects).
  - 7) Serious Treatment-Emergent Adverse Events leading to study discontinuation (number of events, number and percentage of subjects).
  - 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects).

TEAEs will be counted according to the rules below.

### Number of subjects

• Summaries for 2) and 6)

A subject with occurrences of TEAE in both categories (ie, Related and Not Related) will be counted once in the Related category.

Summary for 3)

A subject with an interest of the subject with a subj

Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

Summaries other than 2), 3), and 6)

A subject with multiple occurrences of TEAE will be counted only once.

### Number of events

For each summary, the total number of events will be calculated

7.10.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

Categories:

Intensity

Mild, Moderate, Severe

Time of Onset (day)

[1 - 57, 58 - 169, 170 - 281, 282 - 729, 730 - Max]

Analytical Methods:

The following summaries will be provided using frequency distribution.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Study Treatment-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (6) Intensity of Study Treatment-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (10) Treatment-Emergent Adverse Events of Special Interest by System Organ Class and Preferred Term
- (11) Product Malfunction-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distributions will be provided according to the rules below.

### Number of subjects

• Summary tables other than (5), (6) and (9)

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.

• Summary tables for (5) and (6)

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.

• Summary table for (9)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. Percentages will be based on the number of subjects in the safety analysis set.

7.10.13 Subgroup Analysis of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variables:

**TEAE** 

### Subgroups:

Age  $[Min \le - \le 65, 65 \le - \le Max]$ 

Gender [Male, Female]

Topography of IOs and EOs at Baseline

[1 IO, 2 IOs]

[1 EO, 2 EOs, 3 EOs]

 $[1 EO, 2 \leq EOs]$ 

Previous use of Antibiotics [Yes, No]

Previous use of Immunosuppressants [Yes, No]

Previous use of Biologics [Yes, No]

Concomitant Medications [Biologics only, Immunosuppressants only,

Biologics+Immunosuppressants, None of 2 types of concomitant drugs]

### Analytical Methods:

The following summaries will be provided for each subgroup using frequency distribution. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT.

(1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set for each subgroup.

### 7.10.1.4 Displays of Pretreatment Events

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variables:

 $\mathsf{RTF}$ 

### Analytical Methods:

The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term.
- (2) Serious Pretreatment Events by System Organ Class and Preferred Term.

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

2 Clinical I at

### 7.10.2 Clinical Laboratory Evaluations

7.10.2.1 Hematology and Serum Chemistry

Analysis Set:

Safety Analysis Set

**Analysis Variables:** 

Hematology

Hemoglobin, Hematocrit, Red blood cells count, Mean Corpuscular Volume, Mean Corpuscular Hemoglobin, Mean Corpuscular Hemoglobin Concentration, White blood cells count, differential WBC (Neutrophils, Basophils, Eosinophils, Lymphocytes, Monocytes), Platelet count

Serum Chemistry

C-reactive protein, ALT, AST, Alkaline phosphatase, Gamma-glutamyl transpeptidase, Total bilirubin, Total protein, Glucose, Creatinine, Creatine phosphokinase, Blood urea nitrogen, Potassium, Sodium, Chloride

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 52, Week 104, Week 156 Analytical Methods:

For each variable, summaries (1) to (3) will be provided.

(1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Summary of Shifts of Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

For each laboratory test, the laboratory values will be classified as "Low", "Normal"

only and subject to the applicable Terms of Use or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

### 7.10.2.2 Urinalysis

### Analysis Set:

Safety Analysis Set

### Analysis Variables:

Specific Gravity

рН

[-, +-, +, 2+, 3+]Glucose [-, +-, +, 2+, 3+]Protein [-, +-, +, 2+, 3+]Occult blood [-, +-, +, 2+, 3+]Ketone body [-, +-, +, 2+, 3+]Bilirubin

Urobilinogen [+-, +, 2+, 3+]

### Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 52, Week 104, Week 156 Analytical Methods:

For specific gravity, summaries (1), (2) and (4) will be provided.

For pH, summary (4) will be provided.

For each variable other than specific gravity or pH, summaries (3) and (4) will be provided.

- (1) Summary of Urine Laboratory Test Results and Change from Baseline by Visit Descriptive statistics for observed values for each visit and changes from baseline will be provided.
- (2) Case Plots

Plots over time for each subject will be presented.

(3) Number of Subjects in Categories of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

(4) Summary of Shifts of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

9 May 2022

. A Cach urine laboratory test, the laboratory values will be classified as "Low",
"Normal" or "High" for specific gravity and pH, classified as "Normal" or
"Abnormal" for others relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

al Signs

It:

Analysis Set

triables:

rature

c Blood Pressure

ic Blood Pressure

late

e, Week 2, Week 4, Week 8 Woods 17 was a constant of the provided by the central laboratory. The shift tables will be based on these classifications.

### 7.10.3 Vital Signs

Analysis Set:

Safety Analysis Set

Analysis Variables:

**Temperature** 

Systolic Blood Pressure

Diastolic Blood Pressure

Heart Rate

Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 40, Week 52, Week 78, Week 104, Week 130, Week 156

**Analytical Methods:** 

For each variable, summaries (1) and (2) will be provided

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.

### 7.10.4 Other Observations Related to Safety

7.10.4.1 Donor Specific Antibody

Analysis Set:

Safety Analysis Set

Analysis Variables:

Donor Specific Antibody

[Presence, Absence] (Categories used in analytical methods (1) and (2))

[Presence at baseline and Presence during post-baseline by Week

24,

Presence at baseline and Absence during post-baseline by Week 24,

Absence at baseline and Presence during post-baseline by Week 24,

Absence at baseline and Absence during post-baseline by Week 24]

[Presence at baseline and Presence during post-baseline by Week 52.

Presence at baseline and Absence during post-baseline by Week 52,

Absence at baseline and Presence during post-baseline by Week 52.

Absence at baseline and Absence during post-baseline by Week 52]

[Presence at baseline and Presence during post-baseline by Week 156,

Presence at baseline and Absence during post-baseline by Week 156,

Absence at baseline and Presence during post-baseline by Week 156.

Absence at baseline and Absence during post-baseline by Week 156]

(Categories used in analytical methods (3) and (4))

Property of Lakeda. For hours Presence at baseline and Presence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52 and Presence during post-baseline after Week 52 by Week 156, Presence at baseline and Presence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52 and Absence during post-baseline after Week 52 by Week 156, Presence at baseline and Presence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52 and Presence during post-baseline after Week 52 by Week 156. Presence at baseline and Presence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52 and Absence during post-baseline after Week 52 by Week 156 Presence at baseline and Absence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52 and Presence during post-baseline after Week 52 by Week 156, Presence at baseline and Absence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52 and

Absence during post-baseline after Week 52 by Week 156 Presence at baseline and Absence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52 and Presence during post-baseline after Week 52 by Week 156, Presence at baseline and Absence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52 and Absence during post-baseline after Week 52 by Week 156 Absence at baseline and Presence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52 and Presence during post-baseline after Week 52 by Week 156, Absence at baseline and Presence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52 and Absence during post-baseline after Week 52 by Week 156 Absence at baseline and Presence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52 and Presence during post-baseline after Week 52 by Week 156. Absence at baseline and Presence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52 and and Absence during post-baseline after Week 24 by Week
auting post-baseline after Week 52 by Week 15
and Absence during post-baseline after Week 24 by Week
auting post-baseline after Week 52 by Week 156
Absence at baseline and Absence during post-baseline by V
and Absence during post-baseline after Week 24 by Week 5
Presence during post-baseline after Week 52 by Week 156,
Absence at baseline and Absence during post-baseline by Week 32 by Week 32 by Week 34
Absence during post-baseline after Week 52 by Week 34
Categories used in analytical methods (3)

[Presence during post-baseline by Week 24]

[Presence 3]

[Presence 3] Absence during post-baseline after Week 52 by Week 156 Absence at baseline and Absence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52 and Absence at baseline and Absence during post-baseline by Week 24 and Presence during post-baseline after Week 24 by Week 52 and Absence at baseline and Absence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52 and Absence at baseline and Absence during post-baseline by Week 24 and Absence during post-baseline after Week 24 by Week 52 and

[Presence during post-baseline by Week 24, Absence during post-

[Presence during post-baseline by Week 52, Absence during post-

Presence during post-baseline by Week 156, Absence during post-

[Clearance, non-Clearance]

[Presence at baseline and Clearance, Presence at baseline and non-

Clearance, Absence at baseline and Clearance, Absence at baseline and non-Clearance] (Categories used in analytical method (5))

(Presence/Absence at baseline is results of anti-HLA antibody.)

(Presence/Absence during post-baseline is results of donor specific antibody during post-baseline by Week 24/52/156, ie, Presence if any positive results during post-baseline by Week 24/52/156, Absence if no positive results during post-baseline by Week 24/52/156.)

### Visit:

Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 52, Week 104, Week 156 Analytical Methods:

(1) Summary of Donor Specific Antibody by Visit

Frequency distributions for each visit will be provided

(2) Summary of Shifts of Donor Specific Antibody

Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

(3) Number of Subjects in Categories of Donor Specific Antibody

Frequency distributions of results at baseline and during post-baseline by Week 24/52/156 as well as baseline, during post-baseline by Week 24, during post-baseline after Week 24 by Week 52 and during post-baseline after Week 52 by Week 156 will be provided.

(4) Subgroup Analysis of Efficacy and Safety Endpoints by Donor Specific Antibody

The same analyses of Section 7.8.2.7 and 7.10.1.3 will be conducted for each subgroup of Donor Specific Antibody based on results during post-baseline by Week analyses commission at Week 24

and subgroup of Donor Spec

Week 24/52.

(5) Number of Subjects of Clearance

Frequency distributions of subjects who have assessment

assessment 156. For the same analyses of Section 7.8.2.7, combined remission at Week 24/52, clinical remission at Week 24/52, response at Week 24/52 will be also analyzed for each subgroup of Donor Specific Antibody based on results during post-baseline by

Frequency distributions of results of clearance at Week 156 will be provided for subjects who have presence at any post-baseline visits by Week 104 and have assessment at Week 156. Clearance is defined as the status that subjects have presence at any post-baseline visits by Week 104 with absence at Week 156.

7.10.4.2 Displays of Treatment-Emergent Adverse Events (Japanese)

Analysis Set:

Analysis Variables:

Analytical Methods:

### 7.11

nytical Methods:

TEAEs will be summarized in the same way as in section 7.10.1.2 and 7.10.R.3. All summaries will be presented in Japanese.

Interim Analysis

will not be any interim analysis. Note, the analysis per y analysis for marketing application. Addir:
52 and overall data will be perforively. Just ally sep. A subjects as Plan and September and Septem There will not be any interim analysis. Note, the analysis using data up to Week 24 is the primary analysis for marketing application. Additionally, separate analyses using data up to Week 52 and overall data will be performed after all subjects complete Week 52 and Week 156

### ELECTRONIC SIGNATURES

| | ELECTRONIC SIGNATURES | Z OFFICE |
|---|---|---|
| Signed by | Meaning of Signature | Server Date |
| | Biostatistics Approval | (dd-MMM-yyyy HH;min 'UTC')<br>12-May-2022 01;17 UTC |
| | | 9661 |
| | | "Ve |
| | | 10 |
| | ie | |
| | , slip, | |
| | and | |
| | H | |
| | © 0' | |
| | aicio. | |
| | ane | |
| CO | | |
| 2017 | | |
| LOI' | | |
| ×ô· | | |
| ate. | | |
| lx. | | |
| 100° | | |
| Signed by Signed by Property of Takeda: Property of Takeda: | | |